CLINICAL TRIAL: NCT02064387
Title: A Phase I Open-label, Dose Escalation Study to Investigate the Safety, Pharmacokinetics, Pharmacodynamics, Immunogenicity and Clinical Activity of the Antibody Drug Conjugate GSK2857916 in Subjects With Relapsed/Refractory Multiple Myeloma and Other Advanced Hematologic Malignancies Expressing BCMA
Brief Title: Dose Escalation Study to Investigate the Safety, Pharmacokinetics, Pharmacodynamics, Immunogenicity and Clinical Activity of GSK2857916
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 117159; 2013-004549-18 (EudraCT Number)
Record Dates: First submitted 2014-02-13; First posted 2014-02-17 (Estimated); Results first posted 2019-09-26 (Actual); Last update posted 2020-08-11 (Actual); Status verified 2020-07

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; BCMA expressing Lymphomas
MeSH Terms: conditions — Multiple Myeloma | interventions — belantamab mafodotin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Schedule 1 Part 1 (Experimental): Participants will receive GSK2857916 intravenously over 60 minutes (one dose) every 3 weeks (21 day cycle) for a maximum of 16 cycles.
  Interventions: Drug: GSK2857916
- Schedule 2 Part 1 (Experimental): Participants may receive GSK2857916 intravenously over 60 minutes (one dose) once weekly for three consecutive weeks followed by 1 week of rest (28 day cycle) for a maximum of 16 cycles.
  Interventions: Drug: GSK2857916
- Schedule 1 Part 2 (Experimental): Participants will receive the dose and schedule of GSK2857916 evaluated in Part 1 that is selected for further evaluation in Part 2 for up to 16 cycles.
  Interventions: Drug: GSK2857916
- Schedule 2 Part 2 (Experimental): Participants may receive the dose and schedule of GSK2857916 evaluated in Part 1 that is selected for further evaluation in Part 2 for a maximum of 16 cycles.
  Interventions: Drug: GSK2857916

INTERVENTIONS:
Drug: GSK2857916 — A clear or opalescent solution for IV infusion with unit dose strength of 20 mg/mililiter (mL) for multiple dose levels.

SUMMARY:
This study will assess the safety, pharmacokinetic (PK), pharmacodynamic (PD) and the therapeutic potential of GSK2857916 in subjects with multiple myeloma (MM) and lymphomas that express B cell maturation antigen (BCMA). The hypothesis is that GSK2857916 can be safely administered to subjects with MM and with BCMA positive malignancies at doses where target engagement can be demonstrated. This study will determine if adequate target engagement of BCMA receptors translates into clinical benefit for subjects with MM and BCMA positive lymphomas. The study will consists of two parts: a Part 1 dose escalation phase and a Part 2 expansion phase for safety, tolerability, PK, PD, and clinical activity testing. The study will enroll a total of approximately 80-95 subjects with relapsed/refractory MM or BCMA-expressing hematologic malignancies. The maximum dose to be administered in this trial will not exceed 5 milligram/kilogram(mg/kg).

ELIGIBILITY:
Inclusion Criteria:

* Provide signed written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
* Male or female, 18 years or older (at the time consent is obtained)
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Part 1/dose escalation; Histologically or cytologically confirmed diagnosis of Multiple Myeloma in a subject who fulfills all of the following: has undergone stem cell transplant, or is considered transplant ineligible, has been pretreated with at least the 3 following classes of anti-myeloma drugs: alkylators, proteasome inhibitors and immunomodulators, has demonstrated progression on, or within 60 days of completion of the last therapy.

Part 2 /MM cohort; Histologically or cytologically confirmed diagnosis of: Multiple Myeloma in a subject who fulfills all of the following: has undergone stem cell transplant, or is considered transplant ineligible, has been pretreated with at least the 3 following classes of anti-myeloma drugs: alkylators, proteasome inhibitors and immunomodulators, has demonstrated progression on, or within 60 days of completion of the last therapy, and has measurable disease with at least one of the following: serum M-protein >=0.5 gram (g)/decilitre (dL) (>=5 g/Litre (L)), urine M-protein >=200 milligram (mg)/24hour (h).

Serum free light chain (FLC) assay: Involved FLC level >=5 mg/dL (>=50 mg/L) and an abnormal serum FLC ratio (<0.26 or >1.65) and biopsy proven plasmacytoma (should be measured within 28 days of Screening Visit).

* Part 2/Other BCMA positive Hematologic Malignancies cohort: Subject with one of the following lymphomas: Diffuse Large B-cell Lymphoma (DLBCL) or follicular lymphoma (FL) that exhibits positive BCMA expression on tumor cells as determined by a central laboratory using a validated Immunohistochemistry (IHC) assay. Eligible subjects with BCMA positive malignancies must also fulfill the prior treatment requirements as follows: DLBCL: at least 2 prior lines of systemic therapy containing at least one line of chemo-immunotherapy with anti-CD20 antibody, and either has undergone stem cell transplant or is considered transplant ineligible. FL: at least 2 prior lines of systemic therapy.
* Subjects with a history of autologous stem cell transplant are eligible for study participation provided the following eligibility criteria are met: transplant was > 100 days prior to study enrolment, no active infection; subject meets the remainder of the eligibility criteria outlined in the study protocol.
* Adequate organ system functions as defined below Absolute neutrophil count>=1.0x10^9/L, hemoglobin>=8.0 g/dL, platelet>=50x10^9/L, international normalized ration (INR) <=1.5, Partial thromboplastin time <=1.5xupper limit of normal (ULN), total bilirubin <=1.25xULN, alanine aminotransferase and aspartate aminotransferase<=1.5 X ULN, serum creatinine or calculated creatinine clearance<1.2XULN >=60 mL/min for Part 1;>=50 mL/minute (min) for Part 2 if data supports loosening criteria, Albuminuria<=500 mg/24h, left ventricular ejection fraction >=50%, Troponin<=1xULN, Calcium<=1.1xULN
* A female subject is eligible to participate if she is of: Non-childbearing potential or women of childbearing potential must have a negative serum pregnancy test within 72 hours of first dose of study treatment and agree to use effective contraception during the study and for 60 days following the last dose of study treatment.
* Men with a female partner of childbearing potential must have either had a prior vasectomy or agree to use effective contraception from the time of first dose of study until 60 days after the last dose of study treatment to allow for clearance of any altered sperm
* All prior treatment-related toxicities (defined by National Cancer Institute- Common Toxicity Criteria for Adverse Events, version 4) must be <=Grade 1 at the time of enrollment except for alopecia, and grade 2 neuropathy.

Exclusion Criteria:

* Systemic anti-tumor therapy within 14 days, or plasmapheresis within 7 days prior to the first dose of study drug
* Use of an investigational drug within 14 days or five half-lives, whichever is shorter, preceding the first dose of study drug. Prior treatment with a monoclonal antibody within 30 days of receiving the first dose of study drug.
* History of an allogeneic stem cell transplant. Subjects with a history of an autologous stem cell transplant are NOT excluded if they meet inclusion criteria related to history of autologous stem cell transplant.
* Presence of active renal condition (infection, requirement for dialysis or any other condition that could affect subject's safety). Subjects with isolated proteinuria resulting from MM are eligible, provided they fulfil the inclusion criteria related to organ system function.
* Evidence of active mucosal or internal bleeding
* Any major surgery within the last four weeks.
* Any serious and/or unstable pre-existing medical, psychiatric disorder, or other conditions (including lab abnormalities) that could interfere with subject's safety, obtaining informed consent or compliance to the study procedures.
* Known active infection requiring antibiotic treatment
* Evidence of severe or uncontrolled systemic diseases (e.g., unstable or uncompensated respiratory, hepatic, renal or cardiac disease
* Subjects with previous or concurrent malignancies are allowed only if the second tumor is not contributing to the subject's illness. The subject must not be receiving active therapy, other than hormonal therapy for this disease and the disease must be considered medically stable for at least 2 years.
* Evidence of cardiovascular risk including any of the following: QT interval corrected>=470 millisecond, evidence of current clinically significant uncontrolled arrhythmias, history of myocardial infarction, acute coronary syndromes (including unstable angina), coronary angioplasty, or stenting or bypass grafting within six months of Screening, Class III or IV heart failure as defined by the New York Heart Association functional classification system, uncontrolled hypertension, subjects with intra-cardiac defibrillators or permanent pacemakers, abnormal cardiac valve morphology (>=grade 2) documented by echocardiogram (subjects with grade 1 abnormalities [i.e., mild regurgitation/stenosis] can be entered on study). Subjects with moderate valvular thickening should not be entered on study.
* Known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to GSK2857916 or any of the components of the study treatment.
* Pregnant or lactating female.
* Known human immuno virus infection.
* Subjects with positive test for Hepatitis B surface (HBS-Ag) or Hepatitis B core (HBc)antigen
* Subjects with positive test for hepatitis C (HCV) infection are excluded regardless of viral load. If hepatitis C antibody test is positive, a confirmatory polymerase chain reaction (PCR) or Recombinant immunoblot assay (RIBA) test should be performed. If the PCR or RIBA test is negative, subject is eligible for this trial
* Current active liver or biliary disease (with the exception of Gilbert's syndrome or asymptomatic gallstones, liver metastases or otherwise stable chronic liver disease per investigator's assessment).
* Current corneal disease or a history of corneal disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2014-07-29 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2019-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (9):
- United States (6):
  - GSK Investigational Site, Boston, Massachusetts
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Chapel Hill, North Carolina
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Seattle, Washington
- Canada (2):
  - GSK Investigational Site, Vancouver, British Columbia
  - GSK Investigational Site, Toronto, Ontario
- GSK Investigational Site, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://www.clinicalstudydatarequest.com/SearchAllPostings.aspx?searchparam=117159

REFERENCES:
- [Background] Trudel S, Lendvai N, Popat R, Voorhees PM, Reeves B, Libby EN, Richardson PG, Hoos A, Gupta I, Bragulat V, He Z, Opalinska JB, Cohen AD. Antibody-drug conjugate, GSK2857916, in relapsed/refractory multiple myeloma: an update on safety and efficacy from dose expansion phase I study. Blood Cancer J. 2019 Mar 20;9(4):37. doi: 10.1038/s41408-019-0196-6. PMID 30894515
- [Derived] Collins J, van Noort M, Rathi C, Post TM, Struemper H, Jewell RC, Ferron-Brady G. Longitudinal efficacy and safety modeling and simulation framework to aid dose selection of belantamab mafodotin for patients with multiple myeloma. CPT Pharmacometrics Syst Pharmacol. 2023 Oct;12(10):1411-1424. doi: 10.1002/psp4.13016. Epub 2023 Aug 2. PMID 37465991
- [Derived] Trudel S, Lendvai N, Popat R, Voorhees PM, Reeves B, Libby EN, Richardson PG, Anderson LD Jr, Sutherland HJ, Yong K, Hoos A, Gorczyca MM, Lahiri S, He Z, Austin DJ, Opalinska JB, Cohen AD. Targeting B-cell maturation antigen with GSK2857916 antibody-drug conjugate in relapsed or refractory multiple myeloma (BMA117159): a dose escalation and expansion phase 1 trial. Lancet Oncol. 2018 Dec;19(12):1641-1653. doi: 10.1016/S1470-2045(18)30576-X. Epub 2018 Nov 12. PMID 30442502
- [Derived] Tai YT, Anderson KC. Targeting B-cell maturation antigen in multiple myeloma. Immunotherapy. 2015;7(11):1187-99. doi: 10.2217/imt.15.77. Epub 2015 Sep 15. PMID 26370838

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This is a Phase1 study of antibody drug conjugate GSK2857916 in participants with relapsed/refractory multiple myeloma(MM) or non-hodgkin's lymphoma (NHL).The study was conducted in 2 parts-Part1(dose escalation) and Part2(dose expansion).The starting dose in Part1 was 0.03mg/kg GSK2857916 given once every three weeks; 1cycle=21 days for 16cycles.
Pre-assignment Details: A total of 79 participants were enrolled (38 participants in Part-1 and 41 participants in Part-2).
Groups:
- Part 1: GSK2857916 0.03 mg/kg: Participants were administered a dose of 0.03 milligrams per kilogram (mg/kg) GSK2857916 as intravenous (IV) infusion once every three weeks for a maximum of 16 cycles (1 cycle= 21 days).
- Part 1: GSK2857916 0.06 mg/kg: Participants were administered a dose of 0.06 mg/kg GSK2857916 as IV infusion once every three weeks for a maximum of 16 cycles (1 cycle= 21 days).
- Part 1: GSK2857916 0.12 mg/kg: Participants were administered a dose of 0.12 mg/kg GSK2857916 as IV infusion once every three weeks for a maximum of 16 cycles (1 cycle= 21 days).
- Part 1: GSK2857916 0.24 mg/kg: Participants were administered a dose of 0.24 mg/kg GSK2857916 as IV infusion once every three weeks for a maximum of 16 cycles (1 cycle= 21 days).
- Part 1: GSK2857916 0.48 mg/kg: Participants were administered a dose of 0.48 mg/kg GSK2857916 as IV infusion once every three weeks for a maximum of 16 cycles (1 cycle= 21 days).
- Part 1: GSK2857916 0.96 mg/kg: Participants were administered a dose of 0.96 mg/kg GSK2857916 as IV infusion once every three weeks for a maximum of 16 cycles (1 cycle= 21 days).
- Part 1: GSK2857916 1.92 mg/kg: Participants were administered a dose of 1.92 mg/kg GSK2857916 as IV infusion once every three weeks for a maximum of 16 cycles (1 cycle= 21 days).
- Part 1: GSK2857916 2.50 mg/kg: Participants were administered a dose of 2.50 mg/kg GSK2857916 as IV infusion once every three weeks for a maximum of 16 cycles (1 cycle= 21 days).
- Part 1: GSK2857916 3.40 mg/kg: Participants were administered a dose of 3.40 mg/kg GSK2857916 as IV infusion once every three weeks for a maximum of 16 cycles (1 cycle= 21 days).
- Part 1: GSK2857916 4.60 mg/kg: Participants were administered a dose of 4.60 mg/kg GSK2857916 as IV infusion once every three weeks for a maximum of 16 cycles (1 cycle= 21 days).
- Part 2: GSK2857916 3.40 mg/kg (MM): Participants with multiple myeloma were administered a dose of 3.40 mg/kg GSK2857916 as IV infusion once every three weeks for a maximum of 16 cycles (1 cycle=21 days).
- Part 2: GSK2857916 3.40 mg/kg (NHL): Participants with non-hodgkin's lymphoma were administered a dose of 3.40 mg/kg GSK2857916 as IV infusion once every three weeks for a maximum of 36 cycles (1 cycle=21 days)
Period: Part 1 Max 23.5 Months Followup Duration
Arm/Group | Part 1: GSK2857916 0.03 mg/kg | Part 1: GSK2857916 0.06 mg/kg | Part 1: GSK2857916 0.12 mg/kg | Part 1: GSK2857916 0.24 mg/kg | Part 1: GSK2857916 0.48 mg/kg | Part 1: GSK2857916 0.96 mg/kg | Part 1: GSK2857916 1.92 mg/kg | Part 1: GSK2857916 2.50 mg/kg | Part 1: GSK2857916 3.40 mg/kg | Part 1: GSK2857916 4.60 mg/kg | Part 2: GSK2857916 3.40 mg/kg (MM) | Part 2: GSK2857916 3.40 mg/kg (NHL)
Started | 1 | 1 | 4 | 4 | 4 | 3 | 4 | 8 | 3 | 6 | 0 | 0
Completed | 1 | 1 | 4 | 4 | 4 | 3 | 4 | 6 | 2 | 5 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Period: Part 2 Max 35 Months Followup Duration
Arm/Group | Part 1: GSK2857916 0.03 mg/kg | Part 1: GSK2857916 0.06 mg/kg | Part 1: GSK2857916 0.12 mg/kg | Part 1: GSK2857916 0.24 mg/kg | Part 1: GSK2857916 0.48 mg/kg | Part 1: GSK2857916 0.96 mg/kg | Part 1: GSK2857916 1.92 mg/kg | Part 1: GSK2857916 2.50 mg/kg | Part 1: GSK2857916 3.40 mg/kg | Part 1: GSK2857916 4.60 mg/kg | Part 2: GSK2857916 3.40 mg/kg (MM) | Part 2: GSK2857916 3.40 mg/kg (NHL)
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 35 | 6
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 29 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 3
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 3
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1: GSK2857916 0.03 mg/kg | Part 1: GSK2857916 0.06 mg/kg | Part 1: GSK2857916 0.12 mg/kg | Part 1: GSK2857916 0.24 mg/kg | Part 1: GSK2857916 0.48 mg/kg | Part 1: GSK2857916 0.96 mg/kg | Part 1: GSK2857916 1.92 mg/kg | Part 1: GSK2857916 2.50 mg/kg | Part 1: GSK2857916 3.40 mg/kg | Part 1: GSK2857916 4.60 mg/kg | Part 2: GSK2857916 3.40 mg/kg (MM) | Part 2: GSK2857916 3.40 mg/kg (NHL) | Total
Number analyzed (Participants) | 1 | 1 | 4 | 4 | 4 | 3 | 4 | 8 | 3 | 6 | 35 | 6 | 79
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.0 (NA) — NA indicates that standard deviation could not be calculated for a single participant. | 71.0 (NA) — NA indicates that standard deviation could not be calculated for a single participant. | 56.5 (3.32) | 58.5 (8.35) | 60.0 (10.89) | 58.7 (13.05) | 65.3 (4.79) | 62.6 (11.04) | 48.0 (8.19) | 54.8 (10.11) | 60.5 (7.93) | 60.2 (9.81) | 59.6 (8.90)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 3 | 2 | 2 | 1 | 2 | 5 | 1 | 1 | 18 | 3 | 39
  Male | 0 | 1 | 1 | 2 | 2 | 2 | 2 | 3 | 2 | 5 | 17 | 3 | 40
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Black or African American | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 4 | 0 | 0 | 5 | 0 | 10
  Race: Arabic/North African Heritage | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 2
  Race: White/Caucasian/European Heritage | 1 | 1 | 4 | 3 | 4 | 3 | 3 | 4 | 3 | 5 | 28 | 6 | 65
  Race: Japanese Heritage | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Race: South East Asian Heritage | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Serious Adverse Events (SAEs) and Common (>=5%) Non-serious Adverse Events- Part 1
Description: An adverse event (AE) is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. SAE is defined as any untoward medical occurrence that, at any dose, results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent disability/incapacity, is a congenital anomaly/birth defect, other medical events according to medical or scientific judgement and all events of possible study treatment-induced liver injury with hyperbilirubinemia. Part 1 Population comprised of all Part 1 participants (exclusively MM) who received at least one dose of GSK2857916. SAEs and common (>=5%) non-SAEs is presented.
Time Frame: Up to 23.5 months (maximum duration of follow-up from first dose to last contact or death)
Population: Part 1 Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: GSK2857916 0.03 mg/kg | Part 1: GSK2857916 0.06 mg/kg | Part 1: GSK2857916 0.12 mg/kg | Part 1: GSK2857916 0.24 mg/kg | Part 1: GSK2857916 0.48 mg/kg | Part 1: GSK2857916 0.96 mg/kg | Part 1: GSK2857916 1.92 mg/kg | Part 1: GSK2857916 2.50 mg/kg | Part 1: GSK2857916 3.40 mg/kg | Part 1: GSK2857916 4.60 mg/kg
Number analyzed (Participants) | 1 | 1 | 4 | 4 | 4 | 3 | 4 | 8 | 3 | 6
Participants
  Common non-SAE | 1 | 1 | 4 | 4 | 3 | 3 | 4 | 8 | 3 | 6
  Any SAE | 0 | 0 | 1 | 1 | 1 | 0 | 2 | 4 | 1 | 3

2. Primary Outcome: Number of Participants With SAEs and Common (>=5%) Non-serious Adverse Events- Part 2 (MM)
Description: An adverse event (AE) is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. SAE is defined as any untoward medical occurrence that, at any dose, results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent disability/incapacity, is a congenital anomaly/birth defect, other medical events according to medical or scientific judgement and all events of possible study treatment-induced liver injury with hyperbilirubinemia. Part 2 MM Population comprised of all Part 2 MM participants who received at least one dose of GSK2857916. SAEs and common (>=5%) non-SAEs is presented.
Time Frame: Up to 35 months (maximum duration of follow-up from first dose to last contact or death)
Population: Part 2 MM Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: GSK2857916 3.40 mg/kg (MM)
Number analyzed (Participants) | 35
Participants
  Common non-SAE | 35
  Any SAE | 17

3. Primary Outcome: Number of Participants With SAEs and Common (>=5%) Non-serious Adverse Events- Part 2 (NHL)
Description: An adverse event (AE) is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. SAE is defined as any untoward medical occurrence that, at any dose, results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent disability/incapacity, is a congenital anomaly/birth defect, other medical events according to medical or scientific judgement and all events of possible study treatment-induced liver injury with hyperbilirubinemia. Part 2 NHL Population comprised of all Part 2 NHL participants who received at least one dose of GSK2857916. SAEs and common (>=5%) non-SAEs is presented.
Time Frame: Up to 7.2 months (maximum duration of follow-up from first dose to last contact or death)
Population: Part 2 NHL Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: GSK2857916 3.40 mg/kg (NHL)
Number analyzed (Participants) | 6
Participants
  Common non-SAE | 6
  Any SAE | 3

4. Primary Outcome: Number of Participants With Dose-limiting Toxicities (DLTs) During the Determinative Period- Part 1
Description: An event was considered a DLT if it occurred within the first 21 days of treatment, and met one of the following criteria:albuminuria>=2000mgper24 hour which has been confirmed by repeat test at least7 days apart and is not considered to be related to disease progression, Grade4 neutropenia (without fever) lasting>=7 days, febrile neutropenia lasting>=72 hours, Grade>=3 thrombocytopenia associated with bleeding where estimated blood loss is>10 milliliter orGrade4 thrombocytopenia lasting>7 days and not responding to platelet transfusions, anyGrade3 or greaternon-hematologic toxicity as described in Common National Cancer Institute-Terminology Criteria for Adverse Events version4.0 with the exception of the following Grade3 events that can be controlled within48 hours with routine supportive measures and clinically asymptomatic electrolyte abnormalities which can be corrected within48 hours and liver toxicity meeting pre-specified GSK liver stopping criteria.
Time Frame: Up to Day 21 (from first dose)
Population: DLT Evaluable Population(pop) in Part 1 comprised of All Treated Pop (participants who received at least 1 dose of study treatment) and who received a complete infusion in cycle 1 (once every 3 weeks dosing). Any Part 1 participant in the"All Treated" pop who experiences a DLT, will also be included in the DLT evaluable pop regardless of exposure.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: GSK2857916 0.03 mg/kg | Part 1: GSK2857916 0.06 mg/kg | Part 1: GSK2857916 0.12 mg/kg | Part 1: GSK2857916 0.24 mg/kg | Part 1: GSK2857916 0.48 mg/kg | Part 1: GSK2857916 0.96 mg/kg | Part 1: GSK2857916 1.92 mg/kg | Part 1: GSK2857916 2.50 mg/kg | Part 1: GSK2857916 3.40 mg/kg | Part 1: GSK2857916 4.60 mg/kg
Number analyzed (Participants) | 1 | 1 | 4 | 4 | 4 | 3 | 4 | 8 | 3 | 6
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

5. Primary Outcome: Number of Participants With Grade Change From Baseline in Vital Signs-DBP & SBP-Part 1
Description: Vital signs included systolic blood pressure (SBP), diastolic blood pressure (DBP), temperature (Temp) and heart rate (HR). SBP and DBP were graded using National Cancer Institute-Terminology Criteria for Adverse Events (NCI CTCAE) version 4.0. For SBP: Grade 0-<120 millimeters of mercury[mmHg], 120-139 mmHg[Grade 1], 140-159 mmHg[Grade 2], >=160 mmHg[Grade 3]); For DBP: <80 mmHg [Grade 0], 80-89[Grade 1], 90-99[Grade 2], >=100 mmHg[Grade 3]). An increase is defined as an increase in CTCAE grade relative to Baseline grade. Baseline was defined as the latest pre-dose assessment with a non-missing value, including unscheduled visits. Data for worst-case post Baseline is presented.
Time Frame: Baseline and Up to 21.6 months (maximum duration of follow-up from first dose to last contact or death)
Population: Part 1 Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: GSK2857916 0.03 mg/kg | Part 1: GSK2857916 0.06 mg/kg | Part 1: GSK2857916 0.12 mg/kg | Part 1: GSK2857916 0.24 mg/kg | Part 1: GSK2857916 0.48 mg/kg | Part 1: GSK2857916 0.96 mg/kg | Part 1: GSK2857916 1.92 mg/kg | Part 1: GSK2857916 2.50 mg/kg | Part 1: GSK2857916 3.40 mg/kg | Part 1: GSK2857916 4.60 mg/kg
Number analyzed (Participants) | 1 | 1 | 4 | 4 | 4 | 3 | 4 | 8 | 3 | 6
Participants
  DBP, any grade increase | 0 | 1 | 2 | 1 | 2 | 3 | 3 | 5 | 3 | 4
  SBP, any grade increase | 0 | 1 | 2 | 2 | 3 | 1 | 3 | 7 | 2 | 5

6. Primary Outcome: Number of Participants With Grade Change From Baseline in Vital Signs-DBP & SBP-Part 2 (MM)
Description: Vital signs included SBP, DBP, Temp and HR. SBP and DBP were graded using NCI CTCAE version 4.0. For SBP: Grade 0-<120 mmHg, 120-139 mmHg[Grade 1], 140-159 mmHg[Grade 2], >=160 mmHg[Grade 3]); For DBP: <80 mmHg [Grade 0], 80-89[Grade 1], 90-99[Grade 2], >=100 mmHg[Grade 3]). An increase is defined as an increase in CTCAE grade relative to Baseline grade. Baseline was defined as the latest pre-dose assessment with a non-missing value, including unscheduled visits. Data for worst-case post Baseline is presented.
Time Frame: Baseline and Up to 24.2 months (maximum duration of follow-up from first dose to last contact or death)
Population: Part 2 MM Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: GSK2857916 3.40 mg/kg (MM)
Number analyzed (Participants) | 35
Participants
  DBP, any grade increase | 30
  SBP, any grade increase | 31

7. Primary Outcome: Number of Participants With Grade Change From Baseline in Vital Signs-DBP & SBP-Part 2 (NHL)
Description: Vital signs included SBP, DBP, Temp and HR. SBP and DBP were graded using NCI CTCAE version 4.0. For SBP: Grade 0-<120 mmHg, 120-139 mmHg [Grade 1], 140-159 mmHg[Grade 2], >=160 mmHg [Grade 3]); For DBP: <80 mmHg [Grade 0], 80-89[Grade 1], 90-99[Grade 2], >=100 mmHg[Grade 3]). An increase is defined as an increase in CTCAE grade relative to Baseline grade. Baseline was defined as the latest pre-dose assessment with a non-missing value, including unscheduled visits. Data for worst-case post Baseline is presented.
Time Frame: Up to 7.2 months (maximum duration of follow-up from first dose to last contact or death)
Population: Part 2 NHL Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: GSK2857916 3.40 mg/kg (NHL)
Number analyzed (Participants) | 6
Participants
  DBP, any grade increase | 5
  SBP, any grade increase | 5

8. Primary Outcome: Number of Participants With Change From Baseline in Heart Rate and Temperature-Part 1
Description: The following criteria was used to flag vital signs of potential clinical importance: change from Baseline in heart rate (decrease to <60 beats per minute [bpm] and increase to >100 bpm) and change in temperature from Baseline (increase to >=38 or decrease to <=35 degrees celsius). Baseline was defined as the latest pre-dose assessment with a non-missing value, including unscheduled visits. Data for worst-case post Baseline is presented.
Time Frame: Baseline and Up to 21.6 months (maximum duration of follow-up from first dose to last contact or death)
Population: Part 1 Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: GSK2857916 0.03 mg/kg | Part 1: GSK2857916 0.06 mg/kg | Part 1: GSK2857916 0.12 mg/kg | Part 1: GSK2857916 0.24 mg/kg | Part 1: GSK2857916 0.48 mg/kg | Part 1: GSK2857916 0.96 mg/kg | Part 1: GSK2857916 1.92 mg/kg | Part 1: GSK2857916 2.50 mg/kg | Part 1: GSK2857916 3.40 mg/kg | Part 1: GSK2857916 4.60 mg/kg
Number analyzed (Participants) | 1 | 1 | 4 | 4 | 4 | 3 | 4 | 8 | 3 | 6
Participants
  HR, decrease to <60 | 0 | 0 | 2 | 1 | 0 | 0 | 1 | 4 | 1 | 3
  HR, change to normal or no change | 0 | 0 | 0 | 2 | 1 | 0 | 1 | 3 | 1 | 1
  HR, increase to >100 | 1 | 1 | 2 | 1 | 3 | 3 | 2 | 1 | 1 | 2
  Temp, decrease to <=35 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Temp, change to normal or no change | 1 | 1 | 3 | 4 | 4 | 2 | 4 | 8 | 2 | 6
  Temp, increase to >=38 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0

9. Primary Outcome: Number of Participants With Change From Baseline in Heart Rate and Temperature-Part 2 (MM)
Description: The following criteria was used to flag vital signs of potential clinical importance: change from Baseline in heart rate (decrease to <60 bpm and increase to >100 bpm) and change in temperature from Baseline(increase to >=38 or decrease to <=35 degrees celsius). Baseline was defined as the latest pre-dose assessment with a non-missing value, including unscheduled visits. Data for worst-case post Baseline is presented.
Time Frame: Baseline and Up to 24.2 months (maximum duration of follow-up from first dose to last contact or death)
Population: Part 2 MM Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: GSK2857916 3.40 mg/kg (MM)
Number analyzed (Participants) | 35
Participants
  HR, decrease to <60 | 9
  HR, change to normal or no change | 17
  HR, increase to >100 | 10
  Temp, decrease to <=35 | 1
  Temp, change to normal or no change | 29
  Temp, increase to >=38 | 5

10. Primary Outcome: Number of Participants With Change From Baseline in Heart Rate and Temperature-Part 2 (NHL)
Description: as for outcome 9
Time Frame: Baseline and Up to 7.2 months (maximum duration of follow-up from first dose to last contact or death)
Population: Part 2 NHL Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: GSK2857916 3.40 mg/kg (NHL)
Number analyzed (Participants) | 6
Participants
  HR, decrease to <60 | 3
  HR, change to normal or no change | 2
  HR, increase to >100 | 1
  Temp, decrease to <=35 | 0
  Temp, change to normal or no change | 5
  Temp, increase to >=38 | 1

11. Primary Outcome: Number of Participants With Grade Change From Baseline in Clinical Chemistry Data-Part 1
Description: Blood samples were collected for the analysis of following clinical chemistry parameters: albumin, alkaline phosphatase (ALP), alanine aminotransferase (ALT), aspartate aminotransferase (AST), total bilirubin (T.Bil.), calcium (Ca), creatinine (Creat), creatinine kinase (CK), gamma glutamyl transferase (GGT), glucose (Gl), potassium (Pot), magnesium (Mg), sodium (Sod), phosphate (Ph) and urate. Values(Hyper and hypo)for Gl, Pot, Mg, Sod and Ca is presented. Laboratory parameters were graded according to NCI-CTCAE version 4.0. Grade 1: mild; Grade 2: moderate; Grade 3: severe or medically significant; Grade 4: life-threatening consequences; Grade 5: death related to AE. All increases are an increase in grade from Baseline. Baseline was the latest pre-dose assessment with a non-missing value, including unscheduled visits. Data for worst-case post Baseline is presented.
Time Frame: Baseline and Up to 21.6 months (maximum duration of follow-up from first dose to last contact or death)
Population: Part 1 Population. Only those participants with data available at the specified data points were analyzed (represented by n=X in the category titles).
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: GSK2857916 0.03 mg/kg | Part 1: GSK2857916 0.06 mg/kg | Part 1: GSK2857916 0.12 mg/kg | Part 1: GSK2857916 0.24 mg/kg | Part 1: GSK2857916 0.48 mg/kg | Part 1: GSK2857916 0.96 mg/kg | Part 1: GSK2857916 1.92 mg/kg | Part 1: GSK2857916 2.50 mg/kg | Part 1: GSK2857916 3.40 mg/kg | Part 1: GSK2857916 4.60 mg/kg
Number analyzed (Participants) | 1 | 1 | 4 | 4 | 4 | 3 | 4 | 8 | 3 | 6
Participants
  Gl, Hyper,any grade increase,n=1,1,4,4,4,3,4,8,3,6 | 0 | 0 | 1 | 1 | 4 | 0 | 4 | 6 | 0 | 4
  Gl, Hyper,increase toGrade 3,n=1,1,4,4,4,3,4,8,3,6 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
  Gl, Hyper,increase toGrade 4,n=1,1,4,4,4,3,4,8,3,6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Gl, Hypo,any grade increase,n=1,1,4,4,4,3,4,8,3,6 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 2
  Gl, Hypo,increase toGrade 3,n=1,1,4,4,4,3,4,8,3,6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Gl, Hypo,increase toGrade 4,n=1,1,4,4,4,3,4,8,3,6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Albumin,any grade increase,n=1,1,4,4,4,3,4,8,3,6 | 0 | 0 | 1 | 2 | 3 | 1 | 1 | 1 | 1 | 2
  Albumin,increase to Grade 3,n=1,1,4,4,4,3,4,8,3,6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Albumin,increase to Grade 4,n=1,1,4,4,4,3,4,8,3,6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  ALP,any grade increase,n=1,1,4,4,4,3,4,8,3,6 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 2 | 2 | 5
  ALP,increase to Grade 3,n=1,1,4,4,4,3,4,8,3,6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  ALP,increase to Grade 4,n=1,1,4,4,4,3,4,8,3,6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  ALT,any grade increase,n=1,1,4,4,4,3,4,8,3,6 | 0 | 0 | 1 | 2 | 1 | 0 | 1 | 5 | 1 | 5
  ALT,increase to Grade 3,n=1,1,4,4,4,3,4,8,3,6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  ALT,increase to Grade 4,n=1,1,4,4,4,3,4,8,3,6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  AST,any grade increase,n=1,1,4,4,4,3,4,8,3,6 | 0 | 1 | 2 | 2 | 1 | 1 | 3 | 6 | 3 | 5
  AST,increase to Grade 3,n=1,1,4,4,4,3,4,8,3,6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  AST,increase to Grade 4,n=1,1,4,4,4,3,4,8,3,6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  T.Bil.,any grade increase,n=1,1,4,4,4,3,4,8,3,6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
  T.Bil.,increase to Grade 3,n=1,1,4,4,4,3,4,8,3,6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  T.Bil.,increase to Grade 4,n=1,1,4,4,4,3,4,8,3,6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  CK,any grade increase,n=1,1,4,4,3,3,4,8,3,6: number analyzed (Participants) | 1 | 1 | 4 | 4 | 3 | 3 | 4 | 8 | 3 | 6
  CK,any grade increase,n=1,1,4,4,3,3,4,8,3,6 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 3 | 3 | 3
  CK,increase to Grade 3,n=1,1,4,4,3,3,4,8,3,6: number analyzed (Participants) | 1 | 1 | 4 | 4 | 3 | 3 | 4 | 8 | 3 | 6
  CK,increase to Grade 3,n=1,1,4,4,3,3,4,8,3,6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  CK,increase to Grade 4,n=1,1,4,4,3,3,4,8,3,6: number analyzed (Participants) | 1 | 1 | 4 | 4 | 3 | 3 | 4 | 8 | 3 | 6
  CK,increase to Grade 4,n=1,1,4,4,3,3,4,8,3,6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Creat,any grade increase,n=1,1,4,4,4,3,4,8,3,6 | 0 | 0 | 2 | 0 | 1 | 1 | 1 | 0 | 0 | 0
  Creat,increase to Grade 3,n=1,1,4,4,4,3,4,8,3,6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Creat,increase to Grade 4,n=1,1,4,4,4,3,4,8,3,6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  GGT,any grade increase,1,1,4,4,3,3,4,8,3,6: number analyzed (Participants) | 1 | 1 | 4 | 4 | 3 | 3 | 4 | 8 | 3 | 6
  GGT,any grade increase,1,1,4,4,3,3,4,8,3,6 | 0 | 0 | 1 | 1 | 1 | 0 | 3 | 3 | 3 | 4
  GGT,increase to Grade 3,n=1,1,4,4,3,3,4,8,3,6: number analyzed (Participants) | 1 | 1 | 4 | 4 | 3 | 3 | 4 | 8 | 3 | 6
  GGT,increase to Grade 3,n=1,1,4,4,3,3,4,8,3,6 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
  GGT,increase to Grade 4,n=1,1,4,4,3,3,4,8,3,6: number analyzed (Participants) | 1 | 1 | 4 | 4 | 3 | 3 | 4 | 8 | 3 | 6
  GGT,increase to Grade 4,n=1,1,4,4,3,3,4,8,3,6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Pot,Hyper,any grade increase,n=1,1,4,4,4,3,4,8,3,6 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Pot,Hyper,increase to Grade3,n=1,1,4,4,4,3,4,8,3,6 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Pot,Hyper,increase to Grade4,n=1,1,4,4,4,3,4,8,3,6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Pot,Hypo,any grade increase,n=1,1,4,4,4,3,4,8,3,6 | 0 | 0 | 1 | 1 | 1 | 2 | 0 | 1 | 1 | 2
  Pot,Hypo,increase to Grade3,n=1,1,4,4,4,3,4,8,3,6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Pot,Hypo,increase to Grade4,n=1,1,4,4,4,3,4,8,3,6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Mg,Hyper,any grade increase,n=1,1,4,4,4,3,4,8,3,6 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Mg,Hyper,increase to Grade3,n=1,1,4,4,4,3,4,8,3,6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Mg,Hyper,increase to Grade4,n=1,1,4,4,4,3,4,8,3,6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Mg,Hypo,any grade increase,n=1,1,4,4,4,3,4,8,3,6 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 3 | 0 | 3
  Mg,Hypo,increase to Grade3,n=1,1,4,4,4,3,4,8,3,6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Mg,Hypo,increase to Grade 4,n=1,1,4,4,4,3,4,8,3,6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Ph,any grade increase,n=1,1,4,4,4,3,4,8,3,6 | 0 | 0 | 2 | 1 | 0 | 0 | 1 | 0 | 0 | 0
  Ph,increase to Grade 3,n=1,1,4,4,4,3,4,8,3,6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Ph,increase to Grade 4,n=1,1,4,4,4,3,4,8,3,6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Sod,Hyper,any grade increase,n=1,1,4,4,4,3,4,8,3,6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Sod,Hyper,increase to Grade3,n=1,1,4,4,4,3,4,8,3,6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Sod,Hyper,increase to Grade4,n=1,1,4,4,4,3,4,8,3,6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Sod,Hypo,any grade increase,n=1,1,4,4,4,3,4,8,3,6 | 0 | 1 | 1 | 2 | 2 | 1 | 3 | 2 | 0 | 3
  Sod,Hypo,increase to Grade3,n=1,1,4,4,4,3,4,8,3,6 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2
  Sod,Hypo,increase to Grade4,n=1,1,4,4,4,3,4,8,3,6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Urate,any grade increase,n=1,1,4,4,4,3,4,8,3,6 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Urate,increase to Grade 3,n=1,1,4,4,4,3,4,8,3,6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Urate,increase to Grade4,n=1,1,4,4,4,3,4,8,3,6 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Ca,Hyper,any grade increase,n=1,1,4,4,4,3,4,8,3,6 | 0 | 0 | 1 | 0 | 1 | 1 | 3 | 2 | 0 | 1
  Ca,Hyper,increase to Grade3,n=1,1,4,4,4,3,4,8,3,6 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Ca,Hyper,increase to Grade4,n=1,1,4,4,4,3,4,8,3,6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Ca,Hypo,any grade increase,n=1,1,4,4,4,3,4,8,3,6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1
  Ca,Hypo,increase to Grade3,n=1,1,4,4,4,3,4,8,3,6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Ca,Hypo,increase to Grade4,n=1,1,4,4,4,3,4,8,3,6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

12. Primary Outcome: Number of Participants With Grade Change From Baseline in Clinical Chemistry Data-Part 2 (MM)
Description: Blood samples were collected for the analysis of following clinical chemistry parameters: albumin,ALP,ALT,AST,T.Bil.,Ca, Creat,CK, GGT,Gl, Pot,Mg, Sod, Ph and urate. Values(Hyper and hypo)for Gl, Pot, Mg, Sod and Ca is presented. Laboratory parameters were graded according to NCI-CTCAE version 4.0. Grade 1: mild; Grade 2: moderate; Grade 3: severe or medically significant; Grade 4: life-threatening consequences; Grade 5: death related to AE. All increases are an increase in grade from Baseline. Baseline was the latest pre-dose assessment with a non-missing value, including unscheduled visits. Data for worst-case post Baseline is presented.
Time Frame: Baseline and Up to 24.2 months (maximum duration of follow-up from first dose to last contact or death)
Population: Part 2 MM Population. Only those participants with data available at the specified data points were analyzed (represented by n=X in the category titles).
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: GSK2857916 3.40 mg/kg (MM)
Number analyzed (Participants) | 35
Participants
  Gl, Hyperglycemia,any grade increase,n=35 | 19
  Gl, Hyperglycemia,increase to Grade 3,n=35 | 0
  Gl, Hyperglycemia,increase to Grade 4,n=35 | 0
  Gl, Hypoglycemia,any grade increase,n=35 | 1
  Gl, Hypoglycemia,increase to Grade 3,n=35 | 0
  Gl, Hypoglycemia,increase to Grade 4,n=35 | 0
  Albumin,any grade increase,n=35 | 15
  Albumin,increase to Grade 3,n=35 | 2
  Albumin,increase to Grade 4,n=35 | 0
  ALP,any grade increase,n=35 | 19
  ALP,increase to Grade 3,n=35 | 0
  ALP,increase to Grade 4,,n=35 | 0
  ALT,any grade increase,n=35 | 19
  ALT,increase to Grade 3,n=35 | 0
  ALT,increase to Grade 4,n=35 | 0
  AST,any grade increase,n=35 | 29
  AST,increase to Grade 3,n=35 | 3
  AST,increase to Grade 4,n=35 | 0
  Total bilirubin,any grade increase,n=35 | 3
  Total bilirubin,increase to Grade 3,n=35 | 0
  Total bilirubin,increase to Grade 4,n=35 | 0
  CK,any grade increase,n=35 | 15
  CK,increase to Grade 3,n=35 | 1
  CK,increase to Grade 4 ,n=35 | 0
  Creatinine,any grade increase,n=35 | 7
  Creatinine,increase to Grade 3,n=35 | 0
  Creatinine,increase to Grade 4,n=35 | 0
  GGT,any grade increase,n=34: number analyzed (Participants) | 34
  GGT,any grade increase,n=34 | 21
  GGT,increase to Grade 3,n=34: number analyzed (Participants) | 34
  GGT,increase to Grade 3,n=34 | 6
  GGT,increase to Grade 4,n=34: number analyzed (Participants) | 34
  GGT,increase to Grade 4,n=34 | 0
  Pot,Hyperkalemia,any grade increase,n=35 | 1
  Pot,Hyperkalemia,increase to Grade 3,n=35 | 0
  Pot,Hyperkalemia,increase to Grade 4,n=35 | 1
  Pot,Hypokalemia,any grade increase,n=35 | 12
  Pot,Hypokalemia,increase to Grade 3,n=35 | 3
  Pot,Hypokalemia,increase to Grade 4,n=35 | 1
  Mg,Hypermagnesemia,any grade increase,n=34: number analyzed (Participants) | 34
  Mg,Hypermagnesemia,any grade increase,n=34 | 1
  Mg,Hypermagnesemia,increase to Grade 3,n=34: number analyzed (Participants) | 34
  Mg,Hypermagnesemia,increase to Grade 3,n=34 | 0
  Mg,Hypermagnesemia,increase to Grade 4,n=34: number analyzed (Participants) | 34
  Mg,Hypermagnesemia,increase to Grade 4,n=34 | 0
  Mg,Hypomagnesemia,any grade increase,n=34: number analyzed (Participants) | 34
  Mg,Hypomagnesemia,any grade increase,n=34 | 9
  Mg,Hypomagnesemia,increase to Grade 3,n=34: number analyzed (Participants) | 34
  Mg,Hypomagnesemia,increase to Grade 3,n=34 | 0
  Mg,Hypomagnesemia,increase to Grade 4,n=34: number analyzed (Participants) | 34
  Mg,Hypomagnesemia,increase to Grade 4,n=34 | 1
  Phosphate,any grade increase,n=35 | 8
  Phosphate,increase to Grade 3,n=35 | 0
  Phosphate,increase to Grade 4,n=35 | 0
  Sod,Hypernatremia,any grade increase,n=35 | 0
  Sod,Hypernatremia,increase to Grade 3,n=35 | 0
  Sod,Hypernatremia,increase to Grade 4,n=35 | 0
  Sod,Hyponatremia,any grade increase,n=35 | 4
  Sod,Hyponatremia,increase to Grade 3,n=35 | 0
  Sod,Hyponatremia,increase to Grade 4,n=35 | 1
  Urate,any grade increase,n=35 | 1
  Urate,increase to Grade 3,n=35 | 0
  Urate,increase to Grade 4,n=35 | 1
  Ca,Hypercalcemia,any grade increase,n=35 | 8
  Ca,Hypercalcemia,increase to Grade 3,n=35 | 2
  Ca,Hypercalcemia,increase to Grade 4,,n=35 | 1
  Ca,Hypocalcemia,any grade increase,n=35 | 4
  Ca,Hypocalcemia,increase to Grade 3,n=35 | 0
  Ca,Hypocalcemia,increase to Grade 4,n=35 | 0

13. Primary Outcome: Number of Participants With Grade Change From Baseline in Clinical Chemistry Data-Part 2 (NHL)
Description: Blood samples were collected for the analysis of following clinical chemistry parameters: albumin, ALP, ALT, AST, Bilirubin, Ca, Creat, CK, GGT, Glucose, Pot, Mg, Sod, and Ph. Values(Hyper and hypo)for Glucose, Pot, Mg, Sod and Ca is presented. Laboratory parameters were graded according to NCI-CTCAE version 4.0. Grade 1: mild; Grade 2: moderate; Grade 3: severe or medically significant; Grade 4: life-threatening consequences; Grade 5: death related to AE. All increases are an increase in grade from Baseline. Baseline was the latest pre-dose assessment with a non-missing value, including unscheduled visits. Data for worst-case post Baseline is presented.
Time Frame: Baseline and Up to 7.2 months (maximum duration of follow-up from first dose to last contact or death)
Population: Part 2 NHL Population. Only those participants with data available at the specified data points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: GSK2857916 3.40 mg/kg (NHL)
Number analyzed (Participants) | 5
Participants
  Gl, Hyperglycemia,any grade increase | 2
  Gl, Hyperglycemia,increase to Grade 3 | 0
  Gl, Hyperglycemia,increase to Grade 4 | 0
  Gl, Hypoglycemia,any grade increase | 0
  Gl, Hypoglycemia,increase to Grade 3 | 0
  Gl, Hypoglycemia,increase to Grade 4 | 0
  Albumin,any grade increase | 2
  Albumin,increase to Grade 3 | 0
  Albumin,increase to Grade 4 | 0
  ALP,any grade increase | 1
  ALP,increase to Grade 3 | 0
  ALP,increase to Grade 4 | 0
  ALT,any grade increase | 1
  ALT,increase to Grade 3 | 0
  ALT,increase to Grade 4 | 0
  AST,any grade increase | 2
  AST,increase to Grade 3 | 0
  AST,increase to Grade 4 | 0
  Total bilirubin,any grade increase | 2
  Total bilirubin,increase to Grade 3 | 0
  Total bilirubin,increase to Grade 4 | 0
  CK,any grade increase | 1
  CK,increase to Grade 3 | 0
  CK,increase to Grade 4 | 0
  Creatinine,any grade increase | 1
  Creatinine,increase to Grade 3 | 0
  Creatinine,increase to Grade 4 | 0
  GGT,any grade increase | 2
  GGT,increase to Grade 3 | 0
  GGT,increase to Grade 4 | 0
  Pot,Hyperkalemia,any grade increase | 0
  Pot,Hyperkalemia,increase to Grade 3 | 0
  Pot,Hyperkalemia,increase to Grade 4 | 0
  Pot,Hypokalemia,any grade increase | 1
  Pot,Hypokalemia,increase to Grade 3 | 0
  Pot,Hypokalemia,increase to Grade 4 | 0
  Mg,Hypermagnesemia,any grade increase | 0
  Mg,Hypermagnesemia,increase to Grade 3 | 0
  Mg,Hypermagnesemia,increase to Grade 4 | 0
  Mg,Hypomagnesemia,any grade increase | 1
  Mg,Hypomagnesemia,increase to Grade 3 | 0
  Mg,Hypomagnesemia,increase to Grade 4 | 0
  Phosphate,any grade increase | 2
  Phosphate,increase to Grade 3 | 1
  Phosphate,increase to Grade 4 | 0
  Sod,Hypernatremia,any grade increase | 0
  Sod,Hypernatremia,increase to Grade 3 | 0
  Sod,Hypernatremia,increase to Grade 4 | 0
  Sod,Hyponatremia,any grade increase | 3
  Sod,Hyponatremia,increase to Grade 3 | 0
  Sod,Hyponatremia,increase to Grade 4 | 0
  Ca,Hypercalcemia,any grade increase | 4
  Ca,Hypercalcemia,increase to Grade 3 | 1
  Ca,Hypercalcemia,increase to Grade 4 | 0
  Ca,Hypocalcemia,any grade increase | 1
  Ca,Hypocalcemia,increase to Grade 3 | 0
  Ca,Hypocalcemia,increase to Grade 4 | 0

14. Primary Outcome: Number of Participants With Change From Baseline in Clinical Chemistry Data With Respect to Normal Range-Part 1
Description: Blood samples were collected for the analysis of following clinical chemistry parameters: direct bilirubin (D.Bil.), chloride, carbon dioxide (CO2), lactate dehydrogenase (LDH), total protein (T.Pro) and urea or blood urea nitrogen (BUN). Baseline was defined as latest pre-dose assessment with a non-missing value, including unscheduled visits. A laboratory value that is outside the reference range was considered either high abnormal (value above the upper limit of the reference range) or low abnormal (value below the lower limit of the reference range). If values were unchanged (example: High to High), or whose value became normal, were recorded in the 'To Normal or No Change (NC)' category. Participants were counted twice if the participant "Decreased to low" and "Increased to high" during post-Baseline. Data for worst-case post Baseline is presented.
Time Frame: Baseline and Up to 21.6 months (maximum duration of follow-up from first dose to last contact or death)
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: GSK2857916 0.03 mg/kg | Part 1: GSK2857916 0.06 mg/kg | Part 1: GSK2857916 0.12 mg/kg | Part 1: GSK2857916 0.24 mg/kg | Part 1: GSK2857916 0.48 mg/kg | Part 1: GSK2857916 0.96 mg/kg | Part 1: GSK2857916 1.92 mg/kg | Part 1: GSK2857916 2.50 mg/kg | Part 1: GSK2857916 3.40 mg/kg | Part 1: GSK2857916 4.60 mg/kg
Number analyzed (Participants) | 1 | 1 | 4 | 4 | 4 | 3 | 4 | 8 | 3 | 6
Participants
  D.Bil.,decrease to low,n=1,1,4,2,2,3,4,4,3,5: number analyzed (Participants) | 1 | 1 | 4 | 2 | 2 | 3 | 4 | 4 | 3 | 5
  D.Bil.,decrease to low,n=1,1,4,2,2,3,4,4,3,5 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  D.Bil.,to normal or NC, n=1,1,4,2,2,3,4,4,3,5: number analyzed (Participants) | 1 | 1 | 4 | 2 | 2 | 3 | 4 | 4 | 3 | 5
  D.Bil.,to normal or NC, n=1,1,4,2,2,3,4,4,3,5 | 1 | 1 | 3 | 2 | 1 | 3 | 4 | 3 | 3 | 3
  D.Bil.,increase to high,n=1,1,4,2,2,3,4,4,3,5: number analyzed (Participants) | 1 | 1 | 4 | 2 | 2 | 3 | 4 | 4 | 3 | 5
  D.Bil.,increase to high,n=1,1,4,2,2,3,4,4,3,5 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 2
  Chloride,decrease to low,n=1,1,4,4,4,3,4,8,3,6 | 0 | 0 | 1 | 0 | 2 | 1 | 1 | 3 | 0 | 3
  Chloride,to normal or NC,n=1,1,4,4,4,3,4,8,3,6 | 1 | 1 | 3 | 4 | 2 | 2 | 3 | 4 | 2 | 3
  Chloride,increase to high,n=1,1,4,4,4,3,4,8,3,6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
  CO2,decrease to low,n=1,1,4,4,4,3,4,8,3,6 | 1 | 1 | 1 | 3 | 1 | 1 | 3 | 2 | 2 | 2
  CO2, to normal or NC,n=1,1,4,4,4,3,4,8,3,6 | 0 | 0 | 3 | 1 | 3 | 2 | 0 | 5 | 1 | 4
  CO2,increase to high,n=1,1,4,4,4,3,4,8,3,6 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
  LDH,decrease to low,n=1,1,4,4,3,3,4,8,3,6: number analyzed (Participants) | 1 | 1 | 4 | 4 | 3 | 3 | 4 | 8 | 3 | 6
  LDH,decrease to low,n=1,1,4,4,3,3,4,8,3,6 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
  LDH,to normal or NC,n=n=1,1,4,4,3,3,4,8,3,6: number analyzed (Participants) | 1 | 1 | 4 | 4 | 3 | 3 | 4 | 8 | 3 | 6
  LDH,to normal or NC,n=n=1,1,4,4,3,3,4,8,3,6 | 1 | 1 | 2 | 2 | 1 | 2 | 1 | 5 | 1 | 1
  LDH,increase to high,n=1,1,4,4,3,3,4,8,3,6: number analyzed (Participants) | 1 | 1 | 4 | 4 | 3 | 3 | 4 | 8 | 3 | 6
  LDH,increase to high,n=1,1,4,4,3,3,4,8,3,6 | 0 | 0 | 2 | 1 | 1 | 1 | 3 | 3 | 2 | 5
  T.Pro,decrease to low,n=1,1,4,4,4,3,4,8,3,6 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 2 | 0
  T.Pro,to normal or NC,n=1,1,4,4,4,3,4,8,3,6 | 1 | 1 | 4 | 3 | 2 | 2 | 3 | 6 | 1 | 4
  T.Pro,increase to high,n=1,1,4,4,4,3,4,8,3,6 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 0 | 2
  BUN,decrease to low,n=1,1,4,4,4,3,4,8,3,6 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 1 | 0 | 2
  BUN,to normal or NC,n=1,1,4,4,4,3,4,8,3,6 | 1 | 1 | 2 | 3 | 2 | 3 | 3 | 5 | 2 | 3
  BUN,increase to high,n=1,1,4,4,4,3,4,8,3,6 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 2 | 1 | 1

15. Primary Outcome: Number of Participants With Change From Baseline in Clinical Chemistry Data With Respect to Normal Range-Part 2 (MM)
Description: Blood samples were collected for the analysis of following clinical chemistry parameters: D.Bil., chloride, CO2, LDH, T.Pro and BUN. Baseline was defined as latest pre-dose assessment with a non-missing value, including unscheduled visits.A laboratory value that is outside the reference range was considered either high abnormal (value above the upper limit of the reference range) or low abnormal (value below the lower limit of the reference range). If values were unchanged (example: High to High), or whose value became normal, were recorded in the 'To Normal or NC' category. Participants were counted twice if the participant 'Decreased to Low' and 'Increased to High' during post-Baseline.Data for worst-case post Baseline is presented.
Time Frame: Baseline and Up to 24.2 months (maximum duration of follow-up from first dose to last contact or death)
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: GSK2857916 3.40 mg/kg (MM)
Number analyzed (Participants) | 35
Participants
  D.Bil.,decrease to low,n=30: number analyzed (Participants) | 30
  D.Bil.,decrease to low,n=30 | 2
  D.Bil., to normal or no change,n=30: number analyzed (Participants) | 30
  D.Bil., to normal or no change,n=30 | 20
  D.Bil.,increase to high,n=30: number analyzed (Participants) | 30
  D.Bil.,increase to high,n=30 | 8
  Chloride,decrease to low,n=35 | 7
  Chloride, to normal or no change,n=35 | 25
  Chloride,increase to high,n=35 | 4
  CO2,decrease to low,n=35 | 8
  CO2, to normal or no change,n=35 | 23
  CO2,increase to high,n=35 | 5
  LDH,decrease to low,n=35 | 1
  LDH, to normal or no change,n=35 | 17
  LDH,increase to high,n=35 | 17
  T.Pro,decrease to low,n=35 | 11
  T.Pro, to normal or no change,n=35 | 18
  T.Pro,increase to high,n=35 | 7
  BUN,decrease to low,n=35 | 8
  BUN, to normal or no change,n=35 | 23
  BUN,increase to high,n=35 | 4

16. Primary Outcome: Number of Participants With Change From Baseline in Clinical Chemistry Data With Respect to Normal Range-Part 2 (NHL)
Description: Blood samples were collected for the analysis of following clinical chemistry parameters: D.Bil., chloride, CO2, LDH, and T.Pro. Baseline was defined as latest pre-dose assessment with a non-missing value, including unscheduled visits.A laboratory value that is outside the reference range was considered either high abnormal (value above the upper limit of the reference range) or low abnormal (value below the lower limit of the reference range). If values were unchanged (example: High to High), or whose value became normal, were recorded in the 'To Normal or NC' category. Participants were counted twice if the participant 'Decreased to Low' and 'Increased to High' during post-Baseline. Data for worst-case post Baseline is presented.
Time Frame: Baseline and Up to 7.2 months (maximum duration of follow-up from first dose to last contact or death)
Population: Part 2 NHL Population. Only those participants with data available at the specified data points were analyzed (represented by n=X in the category titles).
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: GSK2857916 3.40 mg/kg (NHL)
Number analyzed (Participants) | 5
Participants
  D.Bil.,decrease to low,n=2: number analyzed (Participants) | 2
  D.Bil.,decrease to low,n=2 | 0
  D.Bil., to normal or no change,n=2: number analyzed (Participants) | 2
  D.Bil., to normal or no change,n=2 | 2
  D.Bil.,increase to high,n=2: number analyzed (Participants) | 2
  D.Bil.,increase to high,n=2 | 0
  Chloride,decrease to low,n=5 | 1
  Chloride, to normal or no change,n=5 | 2
  Chloride,increase to high,n=5 | 2
  CO2,decrease to low,n=5 | 2
  CO2, to normal or no change,n=5 | 3
  CO2,increase to high,n=5 | 0
  LDH,decrease to low,n=5 | 0
  LDH, to normal or no change,n=5 | 4
  LDH,increase to high,n=5 | 1
  T.Pro,decrease to low,n=5 | 1
  T.Pro, to normal or no change,n=5 | 4
  T.Pro,increase to high,n=5 | 0

17. Primary Outcome: Number of Participants With Grade Change From Baseline in Hematology Data-Part 1
Description: Blood samples were collected for the analysis of following hematology parameters: hemoglobin (Hb), lymphocytes (Lymph), neutrophils (Neutro), platelet count (PC), and leukocytes (leuko). The laboratory parameters were graded according to NCI-CTCAE version 4.0. Grade 1: mild; Grade 2: moderate; Grade 3: severe or medically significant; Grade 4: life-threatening consequences; Grade 5: death related to AE. Baseline was defined as latest pre-dose assessment with a non-missing value, including unscheduled visits. An increase is defined as an increase in CTCAE grade relative to Baseline grade. Data for worst-case post Baseline is presented.
Time Frame: Baseline and Up to 21.6 months (maximum duration of follow-up from first dose to last contact or death)
Population: Part 1 Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: GSK2857916 0.03 mg/kg | Part 1: GSK2857916 0.06 mg/kg | Part 1: GSK2857916 0.12 mg/kg | Part 1: GSK2857916 0.24 mg/kg | Part 1: GSK2857916 0.48 mg/kg | Part 1: GSK2857916 0.96 mg/kg | Part 1: GSK2857916 1.92 mg/kg | Part 1: GSK2857916 2.50 mg/kg | Part 1: GSK2857916 3.40 mg/kg | Part 1: GSK2857916 4.60 mg/kg
Number analyzed (Participants) | 1 | 1 | 4 | 4 | 4 | 3 | 4 | 8 | 3 | 6
Participants
  Hb, Hb increased, any grade increase | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Hb, Hb increased, increase to Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hb, Hb increased, increase to Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hb,Anemia, any grade increase | 1 | 1 | 1 | 2 | 2 | 2 | 1 | 3 | 2 | 4
  Hb, Anemia, increase to Grade 3 | 0 | 1 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 1
  Hb, Anemia, increase to Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymph, Lymph count increased, any grade increase | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymph, Lymph count increased, increase to Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymph, Lymph count increased, increase to Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymph, Lymph count decreased, any grade increase | 0 | 0 | 1 | 0 | 2 | 1 | 2 | 4 | 2 | 3
  Lymph, Lymph count decreased, increase to Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 1
  Lymph, Lymph count decreased, increase to Grade 4 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2
  Neutro, any grade increase | 1 | 1 | 2 | 1 | 0 | 2 | 1 | 4 | 2 | 3
  Neutro, increase to Grade 3 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0
  Neutro, increase to Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  PC, any grade increase | 1 | 1 | 2 | 3 | 1 | 1 | 2 | 6 | 3 | 6
  PC, increase to Grade 3 | 1 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 2 | 4
  PC, increase to Grade 4 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Leuko, Leukocytosis, any grade increase | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Leuko, Leukocytosis, increase to Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Leuko, Leukocytosis, increase to Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Leuko, Leuko decreased, any grade increase | 1 | 1 | 3 | 1 | 1 | 1 | 3 | 1 | 2 | 3
  Leuko, Leuko decreased, increase to Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
  Leuko, Leuko decreased, increase to Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

18. Primary Outcome: Number of Participants With Grade Change From Baseline in Hematology Data-Part 2 (MM)
Description: Blood samples were collected for the analysis of following hematology parameters: Hb, Lymph, Neutro, PC, and leuko. The laboratory parameters were graded according to NCI-CTCAE version 4.0. Grade 1: mild; Grade 2: moderate; Grade 3: severe or medically significant; Grade 4: life-threatening consequences; Grade 5: death related to AE. Baseline was defined as the latest pre-dose assessment with a non-missing value, including unscheduled visits.An increase is defined as an increase in CTCAE grade relative to Baseline grade. Data for worst-case post Baseline is presented.
Time Frame: Baseline and Up to 24.2 months (maximum duration of follow-up from first dose to last contact or death)
Population: Part 2 MM Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: GSK2857916 3.40 mg/kg (MM)
Number analyzed (Participants) | 35
Participants
  Hb, Hb increased, any grade increase | 1
  Hb, Hb increased, increase to Grade 3 | 0
  Hb, Hb increased, increase to Grade 4 | 0
  Hb,Anemia, any grade increase | 18
  Hb, Anemia, increase to Grade 3 | 7
  Hb, Anemia, increase to Grade 4 | 0
  Lymph, Lymph count increased, any grade increase | 3
  Lymph, Lymph count increased, increase to Grade 3 | 0
  Lymph, Lymph count increased, increase to Grade 4 | 0
  Lymph, Lymph count decreased, any grade increase | 18
  Lymph, Lymph count decreased, increase to Grade 3 | 8
  Lymph, Lymph count decreased, increase to Grade 4 | 2
  Neutro, any grade increase | 15
  Neutro, increase to Grade 3 | 2
  Neutro, increase to Grade 4 | 5
  PC, any grade increase | 32
  PC, increase to Grade 3 | 13
  PC, increase to Grade 4 | 3
  Leuko, Leukocytosis, any grade increase | 0
  Leuko, Leukocytosis, increase to Grade 3 | 0
  Leuko, Leukocytosis, increase to Grade 4 | 0
  Leuko, Leuko decreased, any grade increase | 16
  Leuko, Leuko decreased, increase to Grade 3 | 4
  Leuko, Leuko decreased, increase to Grade 4 | 1

19. Primary Outcome: Number of Participants With Grade Change From Baseline in Hematology Data-Part 2 (NHL)
Description: Blood samples were collected for the analysis of following hematology parameters: Hb, Lymph, Neutro, PC, and leuko. The laboratory parameters were graded according to NCI-CTCAE version 4.0. Grade 1: mild; Grade 2: moderate; Grade 3: severe or medically significant; Grade 4: life-threatening consequences; Grade 5: death related to AE. Baseline was defined as the latest pre-dose assessment with a non-missing value, including unscheduled visits. An increase is defined as an increase in CTCAE grade relative to Baseline grade. Data for worst-case post Baseline is presented.
Time Frame: Baseline and Up to 7.2 months (maximum duration of follow-up from first dose to last contact or death)
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: GSK2857916 3.40 mg/kg (NHL)
Number analyzed (Participants) | 6
Participants
  Hb, Hb increased, any grade increase, n=6 | 0
  Hb, Hb increased, increase to Grade 3, n=6 | 0
  Hb, Hb increased, increase to Grade 4, n=6 | 0
  Hb,Anemia, any grade increase, n=6 | 2
  Hb, Anemia, increase to Grade 3, n=6 | 0
  Hb, Anemia, increase to Grade 4, n=6 | 0
  Lymph,Lymph count increased,any grade increase,n=6 | 0
  Lymph,Lymph count increased,increase to Grade3,n=6 | 0
  Lymph,Lymph count increased,increase to Grade4,n=6 | 0
  Lymph,Lymph count decreased,any grade increase,n=6 | 5
  Lymph,Lymph count decreased,increase to Grade3,n=6 | 3
  Lymph,Lymph count decreased,increase to Grade4,n=6 | 2
  Neutro, any grade increase, n=6 | 0
  Neutro, increase to Grade 3, n=6 | 0
  Neutro, increase to Grade 4, n=6 | 0
  PC, any grade increase, n=5: number analyzed (Participants) | 5
  PC, any grade increase, n=5 | 3
  PC, increase to Grade 3, n=5: number analyzed (Participants) | 5
  PC, increase to Grade 3, n=5 | 0
  PC, increase to Grade 4, n=5: number analyzed (Participants) | 5
  PC, increase to Grade 4, n=5 | 1
  Leuko, Leukocytosis, any grade increase, n=6 | 0
  Leuko, Leukocytosis, increase to Grade 3, n=6 | 0
  Leuko, Leukocytosis, increase to Grade 4, n=6 | 0
  Leuko, Leuko decreased, any grade increase, n=6 | 4
  Leuko, Leuko decreased, increase to Grade 3, n=6 | 0
  Leuko, Leuko decreased, increase to Grade 4, n=6 | 0

20. Primary Outcome: Number of Participants With Change From Baseline in Hematology Data With Respect to Normal Range-Part 1
Description: Blood samples were collected for the analysis of following hematology parameters: basophils (Baso), eosinophils (Eosino), hematocrit (Hct), mean corpuscular hemoglobin concentration (MCHC), mean corpuscular hemoglobin (MCH), mean corpuscular volume (MCV), monocytes (Mono), erythrocytes (Erythro) and reticulocytes (Reticu). A laboratory value that was outside the reference range was considered either high abnormal (value above the upper limit of the reference range) or low abnormal (value below the lower limit of the reference range). Baseline was defined as latest pre-dose assessment with a non-missing value, including unscheduled visits. If values were unchanged (example: High to High), or whose value became normal, were recorded in the 'To Normal or NC' category. Participants were counted twice if the participant 'Decreased to Low' and 'Increased to High' during post-Baseline.Data at worst-case post Baseline is presented.
Time Frame: Baseline and Up to 21.6 months (maximum duration of follow-up from first dose to last contact or death)
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: GSK2857916 0.03 mg/kg | Part 1: GSK2857916 0.06 mg/kg | Part 1: GSK2857916 0.12 mg/kg | Part 1: GSK2857916 0.24 mg/kg | Part 1: GSK2857916 0.48 mg/kg | Part 1: GSK2857916 0.96 mg/kg | Part 1: GSK2857916 1.92 mg/kg | Part 1: GSK2857916 2.50 mg/kg | Part 1: GSK2857916 3.40 mg/kg | Part 1: GSK2857916 4.60 mg/kg
Number analyzed (Participants) | 1 | 1 | 4 | 4 | 4 | 3 | 4 | 8 | 3 | 6
Participants
  Baso,decrease to low,n=1,1,4,4,4,3,4,8,3,6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
  Baso, to normal or NC,n=1,1,4,4,4,3,4,8,3,6 | 1 | 1 | 4 | 4 | 4 | 3 | 3 | 8 | 3 | 3
  Baso,increase to high,n=1,1,4,4,4,3,4,8,3,6 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 3
  Eosino,decrease to low,n=1,1,4,4,4,3,4,8,3,6 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Eosino,to normal or NC,n=1,1,4,4,4,3,4,8,3,6 | 0 | 1 | 3 | 4 | 4 | 2 | 4 | 8 | 3 | 4
  Eosino,increase to high,n=1,1,4,4,4,3,4,8,3,6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
  Hct,decrease to low,n=1,1,4,4,4,3,4,8,3,6 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 0
  Hct, to normal or NC,n=1,1,4,4,4,3,4,8,3,6 | 1 | 1 | 4 | 3 | 4 | 2 | 4 | 7 | 1 | 6
  Hct,increase to high,n=1,1,4,4,4,3,4,8,3,6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  MCH,decrease to low,n=1,1,4,4,4,3,4,8,3,6 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3 | 1 | 1
  MCH, to normal or NC,n=1,1,4,4,4,3,4,8,3,6 | 1 | 1 | 4 | 4 | 3 | 3 | 1 | 5 | 2 | 5
  MCH,increase to high,n=1,1,4,4,4,3,4,8,3,6 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
  MCHC,decrease to low,n=1,1,4,4,4,3,4,8,3,6 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 3 | 1 | 1
  MCHC, to normal or NC,n=1,1,4,4,4,3,4,8,3,6 | 1 | 0 | 4 | 3 | 4 | 2 | 3 | 5 | 2 | 5
  MCHC,increase to high,n=1,1,4,4,4,3,4,8,3,6 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  MCV,decrease to low,n=1,1,4,4,4,3,4,8,3,6 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 1
  MCV, to normal or NC,n=1,1,4,4,4,3,4,8,3,6 | 1 | 0 | 4 | 4 | 4 | 3 | 2 | 8 | 2 | 5
  MCV,increase to high,n=1,1,4,4,4,3,4,8,3,6 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Mono,decrease to low,n=1,1,4,4,4,3,4,8,3,6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Mono, to normal or NC,n=1,1,4,4,4,3,4,8,3,6 | 0 | 1 | 3 | 3 | 4 | 3 | 2 | 5 | 0 | 1
  Mono,increase to high,n=1,1,4,4,4,3,4,8,3,6 | 1 | 0 | 1 | 1 | 0 | 0 | 2 | 3 | 3 | 5
  Erythro,decrease to low,n=1,1,4,4,4,3,4,8,3,6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
  Erythro, to normal or NC,n=1,1,4,4,4,3,4,8,3,6 | 1 | 1 | 4 | 4 | 4 | 3 | 3 | 6 | 2 | 6
  Erythro,increase to high,n=1,1,4,4,4,3,4,8,3,6 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
  Reticu,decrease to low,n=1,1,3,3,2,1,4,8,2,6: number analyzed (Participants) | 1 | 1 | 3 | 3 | 2 | 1 | 4 | 8 | 2 | 6
  Reticu,decrease to low,n=1,1,3,3,2,1,4,8,2,6 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 3 | 1 | 1
  Reticu,to normal or NC,n=1,1,3,3,2,1,4,8,2,6: number analyzed (Participants) | 1 | 1 | 3 | 3 | 2 | 1 | 4 | 8 | 2 | 6
  Reticu,to normal or NC,n=1,1,3,3,2,1,4,8,2,6 | 1 | 1 | 1 | 3 | 1 | 0 | 1 | 4 | 1 | 4
  Reticu,increase to high,n=1,1,3,3,2,1,4,8,2,6: number analyzed (Participants) | 1 | 1 | 3 | 3 | 2 | 1 | 4 | 8 | 2 | 6
  Reticu,increase to high,n=1,1,3,3,2,1,4,8,2,6 | 0 | 0 | 1 | 0 | 1 | 1 | 3 | 1 | 0 | 1

21. Primary Outcome: Number of Participants With Change From Baseline in Hematology Data With Respect to Normal Range-Part 2 (MM)
Description: Blood samples were collected for the analysis of following hematology parameters: Baso, Eosino, Hct, MCHC, MCH, MCV, Mono, Erythro and Reticu. A laboratory value that was outside the reference range was considered either high abnormal (value above the upper limit of the reference range) or low abnormal (value below the lower limit of the reference range). Baseline was defined as latest pre-dose assessment with a non-missing value, including unscheduled visits. If values were unchanged (example: High to High), or whose value became normal, were recorded in the 'To Normal or NC' category. Participants were counted twice if the participant 'Decreased to Low' and 'Increased to High' during post-Baseline.Data at worst-case post Baseline is presented.
Time Frame: Baseline and Up to 24.2 months (maximum duration of follow-up from first dose to last contact or death)
Population: Part 2 MM Population.Only those participants with data available at the specified data points were analyzed (represented by n=X in the category titles).
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: GSK2857916 3.40 mg/kg (MM)
Number analyzed (Participants) | 35
Participants
  Baso,decrease to low,n=35 | 0
  Baso, to normal or NC,n=35 | 33
  Baso,increase to high,n=35 | 2
  Eosino,decrease to low,n=35 | 7
  Eosino,to normal or NC,n=35 | 26
  Eosino,increase to high,n=35 | 2
  Hct,decrease to low,n=35 | 4
  Hct, to normal or NC,n=35 | 31
  Hct,increase to high,n=35 | 0
  MCH,decrease to low,n=35 | 7
  MCH, to normal or NC,n=35 | 28
  MCH,increase to high,n=35 | 1
  MCHC,decrease to low,n=35 | 5
  MCHC, to normal or NC,n=35 | 28
  MCHC,increase to high,n=35 | 2
  MCV,decrease to low,n=35 | 6
  MCV, to normal or NC,n=35 | 28
  MCV,increase to high,n=35 | 1
  Mono,decrease to low,n=35 | 4
  Mono, to normal or NC,n=35 | 18
  Mono,increase to high,n=35 | 14
  Erythro,decrease to low,n=35 | 2
  Erythro, to normal or NC,n=35 | 31
  Erythro,increase to high,n=35 | 2
  Reticu,decrease to low,n=28: number analyzed (Participants) | 28
  Reticu,decrease to low,n=28 | 10
  Reticu, to normal or NC,n=28: number analyzed (Participants) | 28
  Reticu, to normal or NC,n=28 | 14
  Reticu,increase to high,n=28: number analyzed (Participants) | 28
  Reticu,increase to high,n=28 | 8

22. Primary Outcome: Number of Participants With Change From Baseline in Hematology Data With Respect to Normal Range-Part 2 (NHL)
Description: Blood samples were collected for the analysis of following hematology parameters: Baso, Eosino, Hct, MCHC, MCH, MCV, Mono, Erythro and Reticu. A laboratory value that was outside the reference range was considered either high abnormal (value above the upper limit of the reference range) or low abnormal (value below the lower limit of the reference range). Baseline was defined as latest pre-dose assessment with a non-missing value, including unscheduled visits. If values were unchanged (example: High to High), or whose value became normal, were recorded in the 'To Normal or NC' category. Participants were counted twice if the participant 'Decreased to Low' and 'Increased to High' during post-Baseline. Data at worst-case post Baseline is presented.
Time Frame: Baseline and Up to 7.2 months (maximum duration of follow-up from first dose to last contact or death)
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: GSK2857916 3.40 mg/kg (NHL)
Number analyzed (Participants) | 6
Participants
  Baso,decrease to low,n=6 | 0
  Baso, to normal or NC,n=6 | 6
  Baso,increase to high,n=6 | 0
  Eosino,decrease to low,n=6 | 0
  Eosino,to normal or NC,n=6 | 6
  Eosino,increase to high,n=6 | 0
  Hct,decrease to low,n=6 | 1
  Hct, to normal or NC,n=6 | 5
  Hct,increase to high,n=6 | 0
  MCH,decrease to low,n=6 | 1
  MCH, to normal or NC,n=6 | 5
  MCH,increase to high,n=6 | 0
  MCHC,decrease to low,n=6 | 1
  MCHC, to normal or NC,n=6 | 5
  MCHC,increase to high,n=6 | 0
  MCV,decrease to low,n=6 | 2
  MCV, to normal or NC,n=6 | 4
  MCV,increase to high,n=6 | 0
  Mono,decrease to low,n=6 | 0
  Mono, to normal or NC,n=6 | 4
  Mono,increase to high,n=6 | 2
  Erythro,decrease to low,n=6 | 2
  Erythro, to normal or NC,n=6 | 4
  Erythro,increase to high,n=6 | 0
  Reticu,decrease to low,n=5: number analyzed (Participants) | 5
  Reticu,decrease to low,n=5 | 0
  Reticu, to normal or NC,n=5: number analyzed (Participants) | 5
  Reticu, to normal or NC,n=5 | 4
  Reticu,increase to high,n=5: number analyzed (Participants) | 5
  Reticu,increase to high,n=5 | 1

23. Primary Outcome: Number of Participants With Worst-case Urinalysis Results Post-Baseline Relative to Baseline by Dipstick Method -Part 1
Description: Urine samples were collected to assess urine occult blood (OB) and urine protein (Pro). The dipstick test gave results in a semi-quantitative manner, and results for urinalysis parameters were recorded as no change/decreased, increase to small (indicated by trace and 1+), increase to moderate (indicated by 2+) and increase to large (indicated by 3+ and above) for urine OB and no change/decreased, increase to trace, increase to 1+, increase to 2+ and increase to 3+ for urine Pro indicating proportional concentrations in the urine sample. Baseline was the latest pre-dose assessment with a non-missing value, including unscheduled visits. Data for worst-case post Baseline is presented.
Time Frame: Baseline and Up to 21.6 months (maximum duration of follow-up from first dose to last contact or death)
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: GSK2857916 0.03 mg/kg | Part 1: GSK2857916 0.06 mg/kg | Part 1: GSK2857916 0.12 mg/kg | Part 1: GSK2857916 0.24 mg/kg | Part 1: GSK2857916 0.48 mg/kg | Part 1: GSK2857916 0.96 mg/kg | Part 1: GSK2857916 1.92 mg/kg | Part 1: GSK2857916 2.50 mg/kg | Part 1: GSK2857916 3.40 mg/kg | Part 1: GSK2857916 4.60 mg/kg
Number analyzed (Participants) | 1 | 1 | 4 | 4 | 4 | 3 | 4 | 8 | 3 | 6
Participants
  OB,No change/decreased, n=1,1,4,4,2,3,3,8,3,6: number analyzed (Participants) | 1 | 1 | 4 | 4 | 2 | 3 | 3 | 8 | 3 | 6
  OB,No change/decreased, n=1,1,4,4,2,3,3,8,3,6 | 1 | 1 | 3 | 3 | 1 | 2 | 1 | 5 | 2 | 5
  OB,Increase to small, n=1,1,4,4,2,3,3,8,3,6: number analyzed (Participants) | 1 | 1 | 4 | 4 | 2 | 3 | 3 | 8 | 3 | 6
  OB,Increase to small, n=1,1,4,4,2,3,3,8,3,6 | 0 | 0 | 1 | 0 | 1 | 1 | 2 | 3 | 1 | 0
  OB,Increase to moderate, n=1,1,4,4,2,3,3,8,3,6: number analyzed (Participants) | 1 | 1 | 4 | 4 | 2 | 3 | 3 | 8 | 3 | 6
  OB,Increase to moderate, n=1,1,4,4,2,3,3,8,3,6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  OB,Increase to large, n=1,1,4,4,2,3,3,8,3,6: number analyzed (Participants) | 1 | 1 | 4 | 4 | 2 | 3 | 3 | 8 | 3 | 6
  OB,Increase to large, n=1,1,4,4,2,3,3,8,3,6 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Pro,No change/decreased, n=1,1,4,3,2,3,4,5,3,5: number analyzed (Participants) | 1 | 1 | 4 | 3 | 2 | 3 | 4 | 5 | 3 | 5
  Pro,No change/decreased, n=1,1,4,3,2,3,4,5,3,5 | 1 | 0 | 3 | 3 | 2 | 1 | 3 | 1 | 1 | 1
  Pro,Increase to trace, n=1,1,4,3,2,3,4,5,3,5: number analyzed (Participants) | 1 | 1 | 4 | 3 | 2 | 3 | 4 | 5 | 3 | 5
  Pro,Increase to trace, n=1,1,4,3,2,3,4,5,3,5 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 4 | 2 | 1
  Pro,Increase to 1+, n=1,1,4,3,2,3,4,5,3,5: number analyzed (Participants) | 1 | 1 | 4 | 3 | 2 | 3 | 4 | 5 | 3 | 5
  Pro,Increase to 1+, n=1,1,4,3,2,3,4,5,3,5 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Pro,Increase to 2+, n=1,1,4,3,2,3,4,5,3,5: number analyzed (Participants) | 1 | 1 | 4 | 3 | 2 | 3 | 4 | 5 | 3 | 5
  Pro,Increase to 2+, n=1,1,4,3,2,3,4,5,3,5 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Pro,Increase to 3+, n=1,1,4,3,2,3,4,5,3,5: number analyzed (Participants) | 1 | 1 | 4 | 3 | 2 | 3 | 4 | 5 | 3 | 5
  Pro,Increase to 3+, n=1,1,4,3,2,3,4,5,3,5 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Pro,Unknown, n=1,1,4,3,2,3,4,5,3,5: number analyzed (Participants) | 1 | 1 | 4 | 3 | 2 | 3 | 4 | 5 | 3 | 5
  Pro,Unknown, n=1,1,4,3,2,3,4,5,3,5 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

24. Primary Outcome: Number of Participants With Worst-case Urinalysis Results Post-Baseline Relative to Baseline by Dipstick Method -Part 2 (MM)
Description: Urine samples were collected to assess urine OB and urine Pro. The dipstick test gave results in a semi-quantitative manner, and results for urinalysis parameters were recorded as no change/decreased, increase to small (indicated by trace and 1+), increase to moderate (indicated by 2+) and increase to large (indicated by 3+ and above) for urine OB and no change/decreased, increase to trace, increase to 1+, increase to 2+ and increase to 3+ for urine Pro indicating proportional concentrations in the urine sample. Baseline was the latest pre-dose assessment with a non-missing value, including unscheduled visits. Data for worst-case post Baseline is presented.
Time Frame: Baseline and Up to 24.2 months (maximum duration of follow-up from first dose to last contact or death)
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: GSK2857916 3.40 mg/kg (MM)
Number analyzed (Participants) | 35
Participants
  OB,No change/decreased, n=33: number analyzed (Participants) | 33
  OB,No change/decreased, n=33 | 18
  OB,Increase to small, n=33: number analyzed (Participants) | 33
  OB,Increase to small, n=33 | 14
  OB,Increase to moderate, n=33: number analyzed (Participants) | 33
  OB,Increase to moderate, n=33 | 1
  OB,Increase to large, n=33: number analyzed (Participants) | 33
  OB,Increase to large, n=33 | 0
  Pro,No change/decreased, n=31: number analyzed (Participants) | 31
  Pro,No change/decreased, n=31 | 15
  Pro,Increase to trace, n=31: number analyzed (Participants) | 31
  Pro,Increase to trace, n=31 | 11
  Pro,Increase to 1+, n=31: number analyzed (Participants) | 31
  Pro,Increase to 1+, n=31 | 1
  Pro,Increase to 2+, n=31: number analyzed (Participants) | 31
  Pro,Increase to 2+, n=31 | 0
  Pro,Increase to 3+, n=31: number analyzed (Participants) | 31
  Pro,Increase to 3+, n=31 | 0
  Pro,Unknown, n=31: number analyzed (Participants) | 31
  Pro,Unknown, n=31 | 4

25. Primary Outcome: Number of Participants With Worst-case Urinalysis Results Post-Baseline Relative to Baseline by Dipstick Method -Part 2 (NHL)
Description: Urine samples were collected to assess urine OB and urine Pro. The dipstick test gave results in a semi-quantitative manner, and results for urinalysis parameters were recorded as no change/decreased, increase to small (indicated by trace and 1+), increase to moderate (indicated by 2+) and increase to large (indicated by 3+ and above) for urine OB. For Urine Pro., results were reported as no change/decreased, increase to trace, increase to 1+, increase to 2+ and increase to 3+ indicating proportional concentrations in the urine sample. Baseline was the latest pre-dose assessment with a non-missing value, including unscheduled visits. Data for worst-case post Baseline is presented.
Time Frame: Baseline and Up to 7.2 months (maximum duration of follow-up from first dose to last contact or death)
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: GSK2857916 3.40 mg/kg (NHL)
Number analyzed (Participants) | 5
Participants
  OB,No change/decreased, n=5 | 4
  OB,Increase to small, n=5 | 0
  OB,Increase to moderate, n=5 | 0
  OB,Increase to large, n=5 | 1
  Pro,No change/decreased, n=4: number analyzed (Participants) | 4
  Pro,No change/decreased, n=4 | 3
  Pro,Increase to trace, n=4: number analyzed (Participants) | 4
  Pro,Increase to trace, n=4 | 1
  Pro,Increase to 1+, n=4: number analyzed (Participants) | 4
  Pro,Increase to 1+, n=4 | 0
  Pro,Increase to 2+, n=4: number analyzed (Participants) | 4
  Pro,Increase to 2+, n=4 | 0
  Pro,Increase to 3+, n=4: number analyzed (Participants) | 4
  Pro,Increase to 3+, n=4 | 0

26. Primary Outcome: Change From Baseline in Urine Protein Excretion (24 Hour)-Part 1: GSK2857916 0.06 mg/kg
Description: Urine samples were collected to assess urine Pro. Baseline was the latest pre-dose assessment with a non-missing value, including unscheduled visits. Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value. Data for change from Baseline in urine Pro. excretion (24 hour) is presented
Time Frame: Baseline and Day 1 (Cycle 2 and 3)
Population: Part 1 Population. NA indicates that standard deviation could not be calculated for a single participant.
Measure: Mean (Standard Deviation); unit: Grams per day
Arm/Group | Part 1: GSK2857916 0.06 mg/kg
Number analyzed (Participants) | 1
Grams per day
  Day 1 (Cycle 2) | -0.0 (NA) — NA indicates that standard deviation could not be calculated for a single participant.
  Day 1 (Cycle 3) | 0.3 (NA) — NA indicates that standard deviation could not be calculated for a single participant.

27. Primary Outcome: Change From Baseline in Urine Protein Excretion (24 Hour)-Part 1: GSK2857916 0.03 mg/kg and 0.12 mg/kg
Description: as for outcome 26
Time Frame: Baseline and Day 1 (Cycle 2)
Population: Part 1 Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Grams per day
Arm/Group | Part 1: GSK2857916 0.12 mg/kg | Part 1: GSK2857916 0.03 mg/kg
Number analyzed (Participants) | 3 | 0
Grams per day | 0.4 (0.72) |

28. Primary Outcome: Change From Baseline in Urine Protein Excretion (24 Hour)-Part 1: GSK2857916 0.24 mg/kg
Description: as for outcome 26
Time Frame: Baseline and Day 1 (Cycle 2, 3, 4, 5, 6, 7, 8, 9, 10, 12, 13,14, 15)
Population: Part 1 Population. Only those participants with data available at the specified data points were analyzed. NA indicates that standard deviation could not be calculated for a single participant.
Measure: Mean (Standard Deviation); unit: Grams per day
Arm/Group | Part 1: GSK2857916 0.24 mg/kg
Number analyzed (Participants) | 1
Grams per day
  Day 1 (Cycle 2) | -0.0 (NA) — NA indicates that standard deviation could not be calculated for a single participant.
  Day 1 (Cycle 3) | -0.0 (NA) — NA indicates that standard deviation could not be calculated for a single participant.
  Day 1 (Cycle 4) | 88.1 (NA) — NA indicates that standard deviation could not be calculated for a single participant.
  Day 1 (Cycle 5) | -0.1 (NA) — NA indicates that standard deviation could not be calculated for a single participant.
  Day 1 (Cycle 6) | -0.0 (NA) — NA indicates that standard deviation could not be calculated for a single participant.
  Day 1 (Cycle 7) | -0.0 (NA) — NA indicates that standard deviation could not be calculated for a single participant.
  Day 1 (Cycle 8) | -0.1 (NA) — NA indicates that standard deviation could not be calculated for a single participant.
  Day 1 (Cycle 9) | -0.1 (NA) — NA indicates that standard deviation could not be calculated for a single participant.
  Day 1 (Cycle 10) | -0.1 (NA) — NA indicates that standard deviation could not be calculated for a single participant.
  Day 1 (Cycle 12) | -0.1 (NA) — NA indicates that standard deviation could not be calculated for a single participant.
  Day 1 (Cycle 13) | -0.1 (NA) — NA indicates that standard deviation could not be calculated for a single participant.
  Day 1 (Cycle 14) | -0.1 (NA) — NA indicates that standard deviation could not be calculated for a single participant.
  Day 1 (Cycle 15) | -0.1 (NA) — NA indicates that standard deviation could not be calculated for a single participant.

29. Primary Outcome: Change From Baseline in Urine Protein Excretion (24 Hour)-Part 1: GSK2857916 0.48 mg/kg
Description: as for outcome 26
Time Frame: Baseline and Day 1 (Cycle 2, 3, 5, 6, 7, 8)
Population: Part 1 Population. Only those participants with data available at the specified data points were analyzed (represented by n=X in the category titles). NA indicates that standard deviation could not be calculated for a single participant.
Measure: Mean (Standard Deviation); unit: Grams per day
Arm/Group | Part 1: GSK2857916 0.48 mg/kg
Number analyzed (Participants) | 4
Grams per day
  Day 1 (Cycle 2), n=2: number analyzed (Participants) | 2
  Day 1 (Cycle 2), n=2 | 0.0 (0.04)
  Day 1 (Cycle 3), n=1: number analyzed (Participants) | 1
  Day 1 (Cycle 3), n=1 | 0.8 (NA) — NA indicates that standard deviation could not be calculated for a single participant.
  Day 1 (Cycle 5), n=1: number analyzed (Participants) | 1
  Day 1 (Cycle 5), n=1 | 0.1 (NA) — NA indicates that standard deviation could not be calculated for a single participant.
  Day 1 (Cycle 6), n=1: number analyzed (Participants) | 1
  Day 1 (Cycle 6), n=1 | 0.1 (NA) — NA indicates that standard deviation could not be calculated for a single participant.
  Day 1 (Cycle 7), n=1: number analyzed (Participants) | 1
  Day 1 (Cycle 7), n=1 | 0.1 (NA) — NA indicates that standard deviation could not be calculated for a single participant.
  Day 1 (Cycle 8), n=1: number analyzed (Participants) | 1
  Day 1 (Cycle 8), n=1 | 0.1 (NA) — NA indicates that standard deviation could not be calculated for a single participant.

30. Primary Outcome: Change From Baseline in Urine Protein Excretion (24 Hour)-Part 1: GSK2857916 0.96 mg/kg
Description: as for outcome 26
Time Frame: Baseline and Day 1 (Cycle 2, 3, 4, 5, 6)
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: Grams per day
Arm/Group | Part 1: GSK2857916 0.96 mg/kg
Number analyzed (Participants) | 3
Grams per day
  Day 1 (Cycle 2), n=2: number analyzed (Participants) | 2
  Day 1 (Cycle 2), n=2 | 0.2 (0.35)
  Day 1 (Cycle 3), n=2: number analyzed (Participants) | 2
  Day 1 (Cycle 3), n=2 | -0.1 (0.07)
  Day 1 (Cycle 4), n=1: number analyzed (Participants) | 1
  Day 1 (Cycle 4), n=1 | -0.1 (NA) — NA indicates that standard deviation could not be calculated for a single participant
  Day 1 (Cycle 5), n=1: number analyzed (Participants) | 1
  Day 1 (Cycle 5), n=1 | 0.0 (NA) — NA indicates that standard deviation could not be calculated for a single participant
  Day 1 (Cycle 6), n=1: number analyzed (Participants) | 1
  Day 1 (Cycle 6), n=1 | 0.2 (NA) — NA indicates that standard deviation could not be calculated for a single participant

31. Primary Outcome: Change From Baseline in Urine Protein Excretion (24 Hour)-Part 1: GSK2857916 1.92 mg/kg
Description: as for outcome 26
Time Frame: Baseline and Day 1 (Cycle 2, 3, 4, 5, 6, 7, 8, 11, 12, 13, 14, 16)
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: Grams per day
Arm/Group | Part 1: GSK2857916 1.92 mg/kg
Number analyzed (Participants) | 4
Grams per day
  Day 1 (Cycle 2), n=3: number analyzed (Participants) | 3
  Day 1 (Cycle 2), n=3 | -0.1 (0.48)
  Day 1 (Cycle 3), n=3: number analyzed (Participants) | 3
  Day 1 (Cycle 3), n=3 | -30.3 (51.72)
  Day 1 (Cycle 4), n=4 | -22.4 (45.06)
  Day 1 (Cycle 5), n=3: number analyzed (Participants) | 3
  Day 1 (Cycle 5), n=3 | 0.2 (1.42)
  Day 1 (Cycle 6), n=2: number analyzed (Participants) | 2
  Day 1 (Cycle 6), n=2 | -0.6 (0.99)
  Day 1 (Cycle 7), n=2: number analyzed (Participants) | 2
  Day 1 (Cycle 7), n=2 | -0.6 (1.16)
  Day 1 (Cycle 8), n=2: number analyzed (Participants) | 2
  Day 1 (Cycle 8), n=2 | -0.6 (1.06)
  Day 1 (Cycle 11), n=1: number analyzed (Participants) | 1
  Day 1 (Cycle 11), n=1 | -1.4 (NA) — NA indicates that standard deviation could not be calculated for a single participant.
  Day 1 (Cycle 12), n=1: number analyzed (Participants) | 1
  Day 1 (Cycle 12), n=1 | -1.4 (NA) — NA indicates that standard deviation could not be calculated for a single participant.
  Day 1 (Cycle 13), n=1: number analyzed (Participants) | 1
  Day 1 (Cycle 13), n=1 | -1.4 (NA) — NA indicates that standard deviation could not be calculated for a single participant.
  Day 1 (Cycle 14), n=1: number analyzed (Participants) | 1
  Day 1 (Cycle 14), n=1 | -1.4 (NA) — NA indicates that standard deviation could not be calculated for a single participant.
  Day 1 (Cycle 16), n=1: number analyzed (Participants) | 1
  Day 1 (Cycle 16), n=1 | -1.3 (NA) — NA indicates that standard deviation could not be calculated for a single participant.

32. Primary Outcome: Change From Baseline in Urine Protein Excretion (24 Hour)-Part 1: GSK2857916 2.50 mg/kg
Description: as for outcome 26
Time Frame: Baseline and Day 1 (Cycle 2, 3, 4, 5, 6, 7, 8, 10, 12, 13, 14, 15, 16)
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: Grams per day
Arm/Group | Part 1: GSK2857916 2.50 mg/kg
Number analyzed (Participants) | 8
Grams per day
  Day 1 (Cycle 2), n=4: number analyzed (Participants) | 4
  Day 1 (Cycle 2), n=4 | 0.8 (1.54)
  Day 1 (Cycle 3), n=2: number analyzed (Participants) | 2
  Day 1 (Cycle 3), n=2 | -0.2 (0.31)
  Day 1 (Cycle 4), n=2: number analyzed (Participants) | 2
  Day 1 (Cycle 4), n=2 | -0.2 (0.38)
  Day 1 (Cycle 5), n=1: number analyzed (Participants) | 1
  Day 1 (Cycle 5), n=1 | 0.0 (NA) — NA indicates that standard deviation could not be calculated for a single participant.
  Day 1 (Cycle 6), n=2: number analyzed (Participants) | 2
  Day 1 (Cycle 6), n=2 | -0.2 (0.33)
  Day 1 (Cycle 7), n=1: number analyzed (Participants) | 1
  Day 1 (Cycle 7), n=1 | 0.2 (NA) — NA indicates that standard deviation could not be calculated for a single participant.
  Day 1 (Cycle 8), n=1: number analyzed (Participants) | 1
  Day 1 (Cycle 8), n=1 | -0.5 (NA) — NA indicates that standard deviation could not be calculated for a single participant.
  Day 1 (Cycle 10), n=1: number analyzed (Participants) | 1
  Day 1 (Cycle 10), n=1 | -0.4 (NA) — NA indicates that standard deviation could not be calculated for a single participant.
  Day 1 (Cycle 12), n=1: number analyzed (Participants) | 1
  Day 1 (Cycle 12), n=1 | -0.5 (NA) — NA indicates that standard deviation could not be calculated for a single participant.
  Day 1 (Cycle 13), n=1: number analyzed (Participants) | 1
  Day 1 (Cycle 13), n=1 | -0.5 (NA) — NA indicates that standard deviation could not be calculated for a single participant.
  Day 1 (Cycle 14), n=1: number analyzed (Participants) | 1
  Day 1 (Cycle 14), n=1 | -0.4 (NA) — NA indicates that standard deviation could not be calculated for a single participant.
  Day 1 (Cycle 15), n=1: number analyzed (Participants) | 1
  Day 1 (Cycle 15), n=1 | -0.5 (NA) — NA indicates that standard deviation could not be calculated for a single participant.
  Day 1 (Cycle 16), n=1: number analyzed (Participants) | 1
  Day 1 (Cycle 16), n=1 | -0.5 (NA) — NA indicates that standard deviation could not be calculated for a single participant.

33. Primary Outcome: Change From Baseline in Urine Protein Excretion (24 Hour)-Part 1: GSK2857916 3.40 mg/kg and 4.60 mg/kg
Description: as for outcome 26
Time Frame: Baseline and Day 1 (Cycle 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 15, 16)
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: Grams per day
Arm/Group | Part 1: GSK2857916 3.40 mg/kg | Part 1: GSK2857916 4.60 mg/kg
Number analyzed (Participants) | 3 | 6
Grams per day
  Day 1 (Cycle 2), n=2,5: number analyzed (Participants) | 2 | 5
  Day 1 (Cycle 2), n=2,5 | -0.6 (0.83) | 0.0 (0.45)
  Day 1 (Cycle 3), n=2,4: number analyzed (Participants) | 2 | 4
  Day 1 (Cycle 3), n=2,4 | -0.6 (0.81) | -0.0 (0.23)
  Day 1 (Cycle 4), n=2,4: number analyzed (Participants) | 2 | 4
  Day 1 (Cycle 4), n=2,4 | -0.7 (0.79) | -0.1 (0.25)
  Day 1 (Cycle 5), n=2,4: number analyzed (Participants) | 2 | 4
  Day 1 (Cycle 5), n=2,4 | -0.6 (0.78) | -0.1 (0.46)
  Day 1 (Cycle 6), n=2,4: number analyzed (Participants) | 2 | 4
  Day 1 (Cycle 6), n=2,4 | -0.6 (0.80) | -0.0 (0.33)
  Day 1 (Cycle 7), n=2,4: number analyzed (Participants) | 2 | 4
  Day 1 (Cycle 7), n=2,4 | -0.6 (0.79) | -0.1 (0.48)
  Day 1 (Cycle 8), n=2,2: number analyzed (Participants) | 2 | 2
  Day 1 (Cycle 8), n=2,2 | -0.6 (0.80) | 0.1 (0.15)
  Day 1 (Cycle 9), n=1,2: number analyzed (Participants) | 1 | 2
  Day 1 (Cycle 9), n=1,2 | -1.1 (NA) — NA indicates that standard deviation could not be calculated for a single participant. | 0.2 (0.33)
  Day 1 (Cycle 10), n=1,2: number analyzed (Participants) | 1 | 2
  Day 1 (Cycle 10), n=1,2 | -1.1 (NA) — NA indicates that standard deviation could not be calculated for a single participant. | -0.0 (0.03)
  Day 1 (Cycle 11), n=1,2: number analyzed (Participants) | 1 | 2
  Day 1 (Cycle 11), n=1,2 | -1.2 (NA) — NA indicates that standard deviation could not be calculated for a single participant. | -0.1 (0.06)
  Day 1 (Cycle 12), n=1,2: number analyzed (Participants) | 1 | 2
  Day 1 (Cycle 12), n=1,2 | -1.2 (NA) — NA indicates that standard deviation could not be calculated for a single participant. | 0.0 (0.13)
  Day 1 (Cycle 13), n=1,2: number analyzed (Participants) | 1 | 2
  Day 1 (Cycle 13), n=1,2 | -1.1 (NA) — NA indicates that standard deviation could not be calculated for a single participant. | 0.0 (0.09)
  Day 1 (Cycle 14), n=1,2: number analyzed (Participants) | 1 | 2
  Day 1 (Cycle 14), n=1,2 | -1.0 (NA) — NA indicates that standard deviation could not be calculated for a single participant. | 0.3 (0.11)
  Day 1 (Cycle 15), n=1,2: number analyzed (Participants) | 1 | 2
  Day 1 (Cycle 15), n=1,2 | -1.1 (NA) — NA indicates that standard deviation could not be calculated for a single participant. | 0.1 (0.10)
  Day 1 (Cycle 16), n=1,2: number analyzed (Participants) | 1 | 2
  Day 1 (Cycle 16), n=1,2 | -1.2 (NA) — NA indicates that standard deviation could not be calculated for a single participant. | 0.4 (0.11)

34. Primary Outcome: Change From Baseline in Urine Protein Excretion (24 Hour)-Part 2 (MM)
Description: as for outcome 26
Time Frame: Baseline and Day 1 (Cycle 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 15, 16)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Grams per day
Arm/Group | Part 2: GSK2857916 3.40 mg/kg (MM)
Number analyzed (Participants) | 35
Grams per day
  Day 1 (Cycle 2), n=24: number analyzed (Participants) | 24
  Day 1 (Cycle 2), n=24 | -0.5 (1.21)
  Day 1 (Cycle 3), n=18: number analyzed (Participants) | 18
  Day 1 (Cycle 3), n=18 | -0.7 (1.29)
  Day 1 (Cycle 4), n=13: number analyzed (Participants) | 13
  Day 1 (Cycle 4), n=13 | -0.7 (1.65)
  Day 1 (Cycle 5), n=15: number analyzed (Participants) | 15
  Day 1 (Cycle 5), n=15 | -0.7 (1.66)
  Day 1 (Cycle 6), n=14: number analyzed (Participants) | 14
  Day 1 (Cycle 6), n=14 | -0.8 (1.69)
  Day 1 (Cycle 7), n=14: number analyzed (Participants) | 14
  Day 1 (Cycle 7), n=14 | -0.9 (1.56)
  Day 1 (Cycle 8), n=16: number analyzed (Participants) | 16
  Day 1 (Cycle 8), n=16 | -0.7 (1.53)
  Day 1 (Cycle 9), n=13: number analyzed (Participants) | 13
  Day 1 (Cycle 9), n=13 | -0.5 (1.01)
  Day 1 (Cycle 10), n=12: number analyzed (Participants) | 12
  Day 1 (Cycle 10), n=12 | -0.4 (1.06)
  Day 1 (Cycle 11), n=10: number analyzed (Participants) | 10
  Day 1 (Cycle 11), n=10 | -0.4 (1.01)
  Day 1 (Cycle 12), n=10: number analyzed (Participants) | 10
  Day 1 (Cycle 12), n=10 | -0.4 (1.11)
  Day 1 (Cycle 13), n=9: number analyzed (Participants) | 9
  Day 1 (Cycle 13), n=9 | -0.4 (1.27)
  Day 1 (Cycle 14), n=9: number analyzed (Participants) | 9
  Day 1 (Cycle 14), n=9 | -0.4 (1.25)
  Day 1 (Cycle 15), n=9: number analyzed (Participants) | 9
  Day 1 (Cycle 15), n=9 | -0.4 (1.30)
  Day 1 (Cycle 16), n=9: number analyzed (Participants) | 9
  Day 1 (Cycle 16), n=9 | -0.3 (1.35)

35. Primary Outcome: Change From Baseline in Urine Protein Excretion (24 Hour)-Part 2 (NHL)
Description: Urine samples were collected to assess urine Protein. Baseline was the latest pre-dose assessment with a non-missing value, including unscheduled visits. Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value. Data for change from Baseline in urine Protein excretion (24 hour) is presented.
Time Frame: Baseline and Day 1 (Cycle 2)
Population: Part 2 NHL Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Grams per day
Arm/Group | Part 2: GSK2857916 3.40 mg/kg (NHL)
Number analyzed (Participants) | 2
Grams per day | 0.0 (0.18)

36. Secondary Outcome: Area Under the Concentration-time Curve From Time Zero Extrapolated to Infinite Time (AUC[0-infinity]) of GSK2857916 Following IV Dose in Participants With Relapsed/Refractory MM- Part 1
Description: Blood samples were collected at designated timepoints. Pharmacokinetic (PK) parameters of GSK2857916 were calculated using non-compartmental methods. NA indicates that geometric coefficient of variation could not be calculated for a single participant.
Time Frame: Pre-dose, 30 minutes post start of infusion (SOI), at end of infusion (EOI), 1, 3, 8 and 24 hours post-EOI of Day 1 (Cycle 1)
Population: PK Part 1 Population comprised of Part 1 participants of All Treated Population who had atleast 1 non-missing (non-quantifiable, NQ values were considered non-missing) PK assessment. Only those participants with data available at the specified data points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanogram per milliliter
Arm/Group | Part 1: GSK2857916 0.03 mg/kg | Part 1: GSK2857916 0.06 mg/kg | Part 1: GSK2857916 0.12 mg/kg | Part 1: GSK2857916 0.24 mg/kg | Part 1: GSK2857916 0.48 mg/kg | Part 1: GSK2857916 0.96 mg/kg | Part 1: GSK2857916 1.92 mg/kg | Part 1: GSK2857916 3.40 mg/kg | Part 1: GSK2857916 4.60 mg/kg
Number analyzed (Participants) | 0 | 1 | 4 | 3 | 3 | 2 | 1 | 0 | 4
Hours*nanogram per milliliter |  | 215803.06 (NA) — NA indicates that geometric coefficient of variation could not be calculated for a single participant. | 767285.51 (49.51) | 632339.28 (101.14) | 2991509.97 (72.12) | 9235256.20 (46.65) | 18469186.92 (NA) — NA indicates that geometric coefficient of variation could not be calculated for a single participant. |  | 8355209.26 (25.29)

37. Secondary Outcome: AUC[0-infinity] of GSK2857916 Following IV Dose in Participants With Relapsed/Refractory MM- Part 1: GSK2857916 2.50 mg/kg
Description: Blood samples were collected at designated timepoints. PK parameters of GSK2857916 were calculated using non-compartmental methods.
Time Frame: Pre-dose and EOI of Day 1 (Cycle 1)
Population: PK Part 1 Population. Only those participants with data available at the specified data points were analyzed.
Arm/Group | Part 1: GSK2857916 2.50 mg/kg
Number analyzed (Participants) | 0

38. Secondary Outcome: Area Under the Concentration-time Curve Over the Dosing Interval (AUC[0-tau]) of GSK2857916 Following IV Dose in Participants With Relapsed/Refractory MM- Part 1
Description: Blood samples were collected at designated timepoints. PK parameters of GSK2857916 were calculated using non-compartmental methods. NA indicates that geometric coefficient of variation could not be calculated for a single participant.
Time Frame: Pre-dose, 30 minutes post-SOI, at EOI, 1, 3, 8 and 24 hours post-EOI of Day 1 (Cycle 1)
Population: PK Part 1 Population. Only those participants with data available at the specified data points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanogram per milliliter
Arm/Group | Part 1: GSK2857916 0.03 mg/kg | Part 1: GSK2857916 0.06 mg/kg | Part 1: GSK2857916 0.12 mg/kg | Part 1: GSK2857916 0.24 mg/kg | Part 1: GSK2857916 0.48 mg/kg | Part 1: GSK2857916 0.96 mg/kg | Part 1: GSK2857916 1.92 mg/kg | Part 1: GSK2857916 3.40 mg/kg | Part 1: GSK2857916 4.60 mg/kg
Number analyzed (Participants) | 0 | 1 | 4 | 4 | 3 | 3 | 3 | 2 | 6
Hours*nanogram per milliliter |  | 200467.82 (NA) — NA indicates that geometric coefficient of variation could not be calculated for a single participant. | 633446.78 (35.42) | 729443.84 (91.22) | 2389114.19 (51.12) | 4448319.69 (79.51) | 9892863.42 (51.81) | 23121531.16 (6.59) | 9738914.76 (38.82)

39. Secondary Outcome: AUC[0-tau] of GSK2857916 Following IV Dose in Participants With Relapsed/Refractory MM- Part 1: GSK2857916 2.50 mg/kg
Description: as for outcome 37
Time Frame: Pre-dose and EOI of Day 1 (Cycle 1)
Population: PK Part 1 Population. Only those participants with data available at the specified data points were analyzed.
Arm/Group | Part 1: GSK2857916 2.50 mg/kg
Number analyzed (Participants) | 0

40. Secondary Outcome: Area Under the Concentration-time Curve From Zero to Time of Last Quantifiable Concentration (AUC[0-tlast]) of GSK2857916 Following IV Dose in Participants With Relapsed/Refractory MM- Part 1
Description: as for outcome 38
Time Frame: Pre-dose, 30 minutes post-SOI, at EOI, 1, 3, 8 and 24 hours post-EOI of Day 1 (Cycle 1)
Population: PK Part 1 Population. Only those participants with data available at the specified data points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanogram per milliliter
Arm/Group | Part 1: GSK2857916 0.03 mg/kg | Part 1: GSK2857916 0.06 mg/kg | Part 1: GSK2857916 0.12 mg/kg | Part 1: GSK2857916 0.24 mg/kg | Part 1: GSK2857916 0.48 mg/kg | Part 1: GSK2857916 0.96 mg/kg | Part 1: GSK2857916 1.92 mg/kg | Part 1: GSK2857916 3.40 mg/kg | Part 1: GSK2857916 4.60 mg/kg
Number analyzed (Participants) | 1 | 1 | 4 | 4 | 3 | 3 | 3 | 3 | 6
Hours*nanogram per milliliter | 44260.79 (NA) — NA indicates that geometric coefficient of variation could not be calculated for a single participant. | 178485.20 (NA) — NA indicates that geometric coefficient of variation could not be calculated for a single participant. | 637783.48 (35.67) | 694825.13 (107.50) | 2170746.96 (59.81) | 4492292.65 (82.00) | 10093784.72 (54.20) | 19239850.61 (53.15) | 10131666.86 (47.32)

41. Secondary Outcome: AUC[0-tlast]) of GSK2857916 Following IV Dose in Participants With Relapsed/Refractory MM- Part 1: GSK2857916 2.50 mg/kg
Description: as for outcome 37
Time Frame: Pre-dose and EOI of Day 1 (Cycle 1)
Population: PK Part 1 Population. Only those participants with data available at the specified data points were analyzed.
Arm/Group | Part 1: GSK2857916 2.50 mg/kg
Number analyzed (Participants) | 0

42. Secondary Outcome: Clearance (CL) of GSK2857916 Following IV Dose in Participants With Relapsed/Refractory MM - Part 1
Description: as for outcome 38
Time Frame: Pre-dose, 30 minutes post-SOI, at EOI, 1, 3, 8 and 24 hours post-EOI of Day 1 (Cycle 1)
Population: PK Part 1 Population. Only those participants with data available at the specified data points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Milliliter per hour
Arm/Group | Part 1: GSK2857916 0.03 mg/kg | Part 1: GSK2857916 0.06 mg/kg | Part 1: GSK2857916 0.12 mg/kg | Part 1: GSK2857916 0.24 mg/kg | Part 1: GSK2857916 0.48 mg/kg | Part 1: GSK2857916 0.96 mg/kg | Part 1: GSK2857916 1.92 mg/kg | Part 1: GSK2857916 3.40 mg/kg | Part 1: GSK2857916 4.60 mg/kg
Number analyzed (Participants) | 0 | 1 | 4 | 3 | 3 | 2 | 1 | 0 | 4
Milliliter per hour |  | 28.27 (NA) — NA indicates that geometric coefficient of variation could not be calculated for a single participant. | 10.53 (58.94) | 25.01 (88.61) | 15.10 (75.16) | 8.46 (27.46) | 11.68 (NA) — NA indicates that geometric coefficient of variation could not be calculated for a single participant. |  | 38.84 (37.53)

43. Secondary Outcome: CL of GSK2857916 Following IV Dose in Participants With Relapsed/Refractory MM - Part 1: GSK2857916 2.50 mg/kg
Description: as for outcome 37
Time Frame: Pre-dose and EOI of Day 1 (Cycle 1)
Population: PK Part 1 Population. Only those participants with data available at the specified data points were analyzed.
Arm/Group | Part 1: GSK2857916 2.50 mg/kg
Number analyzed (Participants) | 0

44. Secondary Outcome: Maximum Observed Concentration (Cmax) of GSK2857916 Following IV Dose in Participants With Relapsed/Refractory MM - Part 1
Description: as for outcome 38
Time Frame: Pre-dose, 30 minutes post-SOI, at EOI, 1, 3, 8 and 24 hours post-EOI of Day 1 (Cycle 1)
Population: PK Part 1 Population. Only those participants with data available at the specified data points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per milliliter
Arm/Group | Part 1: GSK2857916 0.03 mg/kg | Part 1: GSK2857916 0.06 mg/kg | Part 1: GSK2857916 0.12 mg/kg | Part 1: GSK2857916 0.24 mg/kg | Part 1: GSK2857916 0.48 mg/kg | Part 1: GSK2857916 0.96 mg/kg | Part 1: GSK2857916 1.92 mg/kg | Part 1: GSK2857916 3.40 mg/kg | Part 1: GSK2857916 4.60 mg/kg
Number analyzed (Participants) | 1 | 1 | 4 | 4 | 3 | 3 | 3 | 3 | 6
Nanograms per milliliter | 429.00 (NA) — NA indicates that geometric coefficient of variation could not be calculated for a single participant. | 1323.00 (NA) — NA indicates that geometric coefficient of variation could not be calculated for a single participant. | 2956.77 (18.45) | 4548.10 (20.27) | 11876.46 (24.08) | 23050.05 (23.05) | 43774.18 (45.18) | 68128.02 (20.84) | 117385.57 (24.14)

45. Secondary Outcome: Cmax of GSK2857916 Following IV Dose in Participants With Relapsed/Refractory MM - Part 1: GSK2857916 2.50 mg/kg
Description: as for outcome 37
Time Frame: Pre-dose and EOI of Day 1 (Cycle 1)
Population: PK Part 1 Population. Only those participants with data available at the specified data points were analyzed.
Arm/Group | Part 1: GSK2857916 2.50 mg/kg
Number analyzed (Participants) | 0

46. Secondary Outcome: Trough Plasma Concentration (Ctrough) of GSK2857916 Following IV Dose in Participants With Relapsed/Refractory MM - Part 1
Description: Blood samples were collected at designated timepoints. PK parameters of GSK2857916 were calculated using non-compartmental methods. NA indicates that the geometric mean and geometric coefficient of variation could not be calculated since the concentration was not quantifiable. NA indicates that geometric coefficient of variation could not be calculated for a single participant.
Time Frame: Pre-dose, 30 minutes post-SOI, at EOI, 1, 3, 8 and 24 hours post-EOI of Day 1 (Cycle 1), Pre-dose and EOI of Day 1 (Cycle 2 and Cycle 4)
Population: PK Part 1 Population. Only those participants with data available at the specified data points were analyzed (represented by n=X in the category titles).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per milliliter
Arm/Group | Part 1: GSK2857916 0.03 mg/kg | Part 1: GSK2857916 0.06 mg/kg | Part 1: GSK2857916 0.12 mg/kg | Part 1: GSK2857916 0.24 mg/kg | Part 1: GSK2857916 0.48 mg/kg | Part 1: GSK2857916 0.96 mg/kg | Part 1: GSK2857916 1.92 mg/kg | Part 1: GSK2857916 3.40 mg/kg | Part 1: GSK2857916 4.60 mg/kg
Number analyzed (Participants) | 1 | 1 | 4 | 4 | 4 | 3 | 4 | 3 | 6
Nanograms per milliliter
  Day 1, Cycle 1,n=0,1,4,2,1,3,3,2,6: number analyzed (Participants) | 0 | 1 | 4 | 2 | 1 | 3 | 3 | 2 | 6
  Day 1, Cycle 1,n=0,1,4,2,1,3,3,2,6 |  | NA (NA) — NA indicates that the geometric mean and geometric coefficient of variation could not be calculated since the concentration was not quantifiable. | 381.95 (105.55) | 1331.11 (44.43) | 4307.00 (NA) — NA indicates that geometric coefficient of variation could not be calculated for a single participant. | 3720.27 (113.71) | 11420.61 (35.70) | 28134.46 (35.97) | 2301.18 (75.69)
  Day 1, Cycle 2,n=0,1,0,2,1,2,2,2,5: number analyzed (Participants) | 0 | 1 | 0 | 2 | 1 | 2 | 2 | 2 | 5
  Day 1, Cycle 2,n=0,1,0,2,1,2,2,2,5 |  | NA (NA) — NA indicates that the geometric mean and geometric coefficient of variation could not be calculated since the concentration was not quantifiable. |  | 1672.18 (28.76) | 7259.00 (NA) — NA indicates that geometric coefficient of variation could not be calculated for a single participant. | 9510.04 (104.56) | 12791.83 (46.82) | 12719.77 (6.21) | 2643.94 (123.56)
  Day 1, Cycle 4,n=0,0,0,0,0,0,0,0,0: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

47. Secondary Outcome: Ctrough of GSK2857916 Following IV Dose in Participants With Relapsed/Refractory MM - Part 1: GSK2857916 2.50 mg/kg
Description: as for outcome 37
Time Frame: Pre-dose and EOI of Day 1 (Cycle 1, Cycle 2 and Cycle 4)
Population: PK Part 1 Population.Only those participants with data available at the specified data points were analyzed (represented by n=X in the category titles).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per milliliter
Arm/Group | Part 1: GSK2857916 2.50 mg/kg
Number analyzed (Participants) | 8
Nanograms per milliliter
  Day 1, Cycle 1,n=8 | 3726.78 (49.92)
  Day 1, Cycle 2,n=4: number analyzed (Participants) | 4
  Day 1, Cycle 2,n=4 | 11352.94 (268.64)
  Day 1, Cycle 4,n=3: number analyzed (Participants) | 3
  Day 1, Cycle 4,n=3 | 11121.73 (59.75)

48. Secondary Outcome: Terminal Half-life (t1/2) of GSK2857916 Following IV Dose in Participants With Relapsed/Refractory MM - Part 1
Description: as for outcome 38
Time Frame: Pre-dose, 30 minutes post-SOI, at EOI, 1, 3, 8 and 24 hours post-EOI of Day 1 (Cycle 1)
Population: PK Part 1 Population. Only those participants with data available at the specified data points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Part 1: GSK2857916 0.03 mg/kg | Part 1: GSK2857916 0.06 mg/kg | Part 1: GSK2857916 0.12 mg/kg | Part 1: GSK2857916 0.24 mg/kg | Part 1: GSK2857916 0.48 mg/kg | Part 1: GSK2857916 0.96 mg/kg | Part 1: GSK2857916 1.92 mg/kg | Part 1: GSK2857916 3.40 mg/kg | Part 1: GSK2857916 4.60 mg/kg
Number analyzed (Participants) | 0 | 1 | 4 | 3 | 3 | 2 | 1 | 0 | 4
Hours |  | 126.18 (NA) — NA indicates that geometric coefficient of variation could not be calculated for a single participant. | 188.20 (37.41) | 117.82 (76.00) | 198.48 (50.42) | 264.93 (46.73) | 308.39 (NA) — NA indicates that geometric coefficient of variation could not be calculated for a single participant. |  | 103.74 (17.29)

49. Secondary Outcome: t1/2 of GSK2857916 Following IV Dose in Participants With Relapsed/Refractory MM - Part 1: GSK2857916 2.50 mg/kg
Description: as for outcome 37
Time Frame: Pre-dose and EOI of Day 1 (Cycle 1)
Population: PK Part 1 Population. Only those participants with data available at the specified data points were analyzed.
Arm/Group | Part 1: GSK2857916 2.50 mg/kg
Number analyzed (Participants) | 0

50. Secondary Outcome: Volume of Distribution at Steady State (Vss) of GSK2857916 Following IV Dose in Participants With Relapsed/Refractory MM - Part 1
Description: as for outcome 38
Time Frame: Pre-dose, 30 minutes post-SOI, at EOI, 1, 3, 8 and 24 hours post-EOI of Day 1 (Cycle 1)
Population: PK Part 1 Population. Only those participants with data available at the specified data points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Milliliter
Arm/Group | Part 1: GSK2857916 0.03 mg/kg | Part 1: GSK2857916 0.06 mg/kg | Part 1: GSK2857916 0.12 mg/kg | Part 1: GSK2857916 0.24 mg/kg | Part 1: GSK2857916 0.48 mg/kg | Part 1: GSK2857916 0.96 mg/kg | Part 1: GSK2857916 1.92 mg/kg | Part 1: GSK2857916 3.40 mg/kg | Part 1: GSK2857916 4.60 mg/kg
Number analyzed (Participants) | 0 | 1 | 4 | 3 | 3 | 2 | 1 | 0 | 4
Milliliter |  | 5239 (NA) — NA indicates that geometric coefficient of variation could not be calculated for a single participant. | 2900 (29.04) | 4286 (31.29) | 4388 (21.99) | 3224 (22.37) | 5156 (NA) — NA indicates that geometric coefficient of variation could not be calculated for a single participant. |  | 5215 (19.41)

51. Secondary Outcome: Vss of GSK2857916 Following IV Dose in Participants With Relapsed/Refractory MM - Part 1: GSK2857916 2.50 mg/kg
Description: as for outcome 37
Time Frame: Pre-dose and EOI of Day 1 (Cycle 1)
Population: PK Part 1 Population. Only those participants with data available at the specified data points were analyzed.
Arm/Group | Part 1: GSK2857916 2.50 mg/kg
Number analyzed (Participants) | 0

52. Secondary Outcome: Time to Reach Maximum Observed Concentration (Tmax) of GSK2857916 Following IV Dose in Participants With Relapsed/Refractory MM - Part 1
Description: Blood samples were collected at designated timepoints. PK parameters of GSK2857916 were calculated using non-compartmental methods. Median and full range of Tmax have been presented.
Time Frame: Pre-dose, 30 minutes post-SOI, at EOI, 1, 3, 8 and 24 hours post-EOI of Day 1 (Cycle 1)
Population: PK Part 1 Population. Only those participants with data available at the specified data points were analyzed.
Measure: Median (Full Range); unit: Hours
Arm/Group | Part 1: GSK2857916 0.03 mg/kg | Part 1: GSK2857916 0.06 mg/kg | Part 1: GSK2857916 0.12 mg/kg | Part 1: GSK2857916 0.24 mg/kg | Part 1: GSK2857916 0.48 mg/kg | Part 1: GSK2857916 0.96 mg/kg | Part 1: GSK2857916 1.92 mg/kg | Part 1: GSK2857916 3.40 mg/kg | Part 1: GSK2857916 4.60 mg/kg
Number analyzed (Participants) | 1 | 1 | 4 | 4 | 3 | 3 | 3 | 3 | 6
Hours | 2.080 [2.08 to 2.08] | 4.080 [4.08 to 4.08] | 1.185 [1.00 to 2.00] | 3.085 [2.00 to 8.78] | 1.000 [1.00 to 4.00] | 2.050 [2.00 to 2.08] | 1.000 [0.50 to 24.00] | 6.920 [2.02 to 8.78] | 1.560 [0.95 to 2.07]

53. Secondary Outcome: Tmax of GSK2857916 Following IV Dose in Participants With Relapsed/Refractory MM - Part 1: GSK2857916 2.50 mg/kg
Description: as for outcome 52
Time Frame: Pre-dose and EOI of Day 1 (Cycle 1)
Population: PK Part 1 Population. Only those participants with data available at the specified data points were analyzed.
Arm/Group | Part 1: GSK2857916 2.50 mg/kg
Number analyzed (Participants) | 0

54. Secondary Outcome: Ctrough of GSK2857916 Following IV Dose in Participants With Relapsed/Refractory MM-Part 2
Description: as for outcome 37
Time Frame: Pre-dose and EOI of Day 1 (Cycle 1, Cycle 2 and Cycle 4)
Population: PK Part 2 MM Population comprised of Part 2 MM participants of All Treated Population who had atleast 1 non-missing (NQ) PK assessment. Only those participants with data available at the specified data points were analyzed (represented by n=X in the category titles).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per milliliter
Arm/Group | Part 2: GSK2857916 3.40 mg/kg (MM)
Number analyzed (Participants) | 35
Nanograms per milliliter
  Day 1, Cycle 1,n=28: number analyzed (Participants) | 28
  Day 1, Cycle 1,n=28 | 3486.49 (85.71)
  Day 1, Cycle 2,n=18: number analyzed (Participants) | 18
  Day 1, Cycle 2,n=18 | 5799.89 (66.52)
  Day 1, Cycle 4,n=12: number analyzed (Participants) | 12
  Day 1, Cycle 4,n=12 | 6184.46 (103.79)

55. Secondary Outcome: Ctrough of GSK2857916 Following IV Dose in Participants With NHL-Part 2
Description: as for outcome 37
Time Frame: Pre-dose and EOI of Day 1 (Cycle 1, Cycle 2 and Cycle 3)
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: Nanograms per milliliter
Arm/Group | Part 2: GSK2857916 3.40 mg/kg (NHL)
Number analyzed (Participants) | 5
Nanograms per milliliter
  Cycle 1 Day 1, n=5 | 0.0 (0.00)
  Cycle 2 Day 1, n=4: number analyzed (Participants) | 4
  Cycle 2 Day 1, n=4 | 3761.8 (2225.57)
  Cycle 3 Day 1, n=1: number analyzed (Participants) | 1
  Cycle 3 Day 1, n=1 | 8401.0 (NA) — NA indicates that standard deviation could not be calculated for a single participant.

56. Secondary Outcome: AUC(0-tlast) of Cys Monomethyl Auristatin F (Cys-mcMMAF) Following IV Dose of GSK2857916 in Participants With Relapsed/Refractory MM- Part 1
Description: Blood samples were collected at designated timepoints. PK parameters of Cys-mcMMAF were calculated using non-compartmental methods. NA indicates that geometric coefficient of variation could not be calculated for a single participant.
Time Frame: Pre-dose, 30 minutes post-SOI, at EOI, 1, 3, 8 and 24 hours post-EOI of Day 1 (Cycle 1)
Population: PK Part 1 Population. Only those participants with data available at the specified data points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*picogram per milliliter
Arm/Group | Part 1: GSK2857916 0.03 mg/kg | Part 1: GSK2857916 0.06 mg/kg | Part 1: GSK2857916 0.12 mg/kg | Part 1: GSK2857916 0.24 mg/kg | Part 1: GSK2857916 0.48 mg/kg | Part 1: GSK2857916 0.96 mg/kg | Part 1: GSK2857916 1.92 mg/kg | Part 1: GSK2857916 3.40 mg/kg | Part 1: GSK2857916 4.60 mg/kg
Number analyzed (Participants) | 0 | 0 | 1 | 4 | 3 | 3 | 3 | 3 | 6
Hours*picogram per milliliter |  |  | 1157.46 (NA) — NA indicates that geometric coefficient of variation could not be calculated for a single participant. | 1623.87 (41.43) | 14681.62 (91.88) | 20787.48 (209.27) | 72608.00 (17.60) | 119177.30 (35.77) | 181147.61 (94.32)

57. Secondary Outcome: AUC(0-tlast) of Cys-mcMMAF Following IV Dose of GSK2857916 in Participants With Relapsed/Refractory MM- Part 1: GSK2857916 2.50 mg/kg
Description: Blood samples were collected at designated timepoints. PK parameters of Cys-mcMMAF were calculated using non-compartmental methods.
Time Frame: Pre-dose and EOI of Day 1 (Cycle 1)
Population: PK Part 1 Population. Only those participants with data available at the specified data points were analyzed.
Arm/Group | Part 1: GSK2857916 2.50 mg/kg
Number analyzed (Participants) | 0

58. Secondary Outcome: Cmax of Cys-mcMMAF Following IV Dose of GSK2857916 in Participants With Relapsed/Refractory MM- Part 1
Description: as for outcome 56
Time Frame: Pre-dose, 30 minutes post-SOI, at EOI, 1, 3, 8 and 24 hours post-EOI of Day 1 (Cycle 1)
Population: PK Part 1 Population. Only those participants with data available at the specified data points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Picograms per milliliter
Arm/Group | Part 1: GSK2857916 0.03 mg/kg | Part 1: GSK2857916 0.06 mg/kg | Part 1: GSK2857916 0.12 mg/kg | Part 1: GSK2857916 0.24 mg/kg | Part 1: GSK2857916 0.48 mg/kg | Part 1: GSK2857916 0.96 mg/kg | Part 1: GSK2857916 1.92 mg/kg | Part 1: GSK2857916 3.40 mg/kg | Part 1: GSK2857916 4.60 mg/kg
Number analyzed (Participants) | 0 | 0 | 1 | 4 | 3 | 3 | 3 | 3 | 6
Picograms per milliliter |  |  | 51.50 (NA) — NA indicates that geometric coefficient of variation could not be calculated for a single participant. | 91.49 (31.76) | 260.62 (15.70) | 488.29 (38.51) | 1054.02 (18.96) | 1199.86 (35.11) | 2544.02 (87.04)

59. Secondary Outcome: Cmax of Cys-mcMMAF Following IV Dose of GSK2857916 in Participants With Relapsed/Refractory MM- Part 1: GSK2857916 2.50 mg/kg
Description: as for outcome 57
Time Frame: Pre-dose and EOI of Day 1 (Cycle 1)
Population: PK Part 1 Population. Only those participants with data available at the specified data points were analyzed.
Arm/Group | Part 1: GSK2857916 2.50 mg/kg
Number analyzed (Participants) | 0

60. Secondary Outcome: Ctrough of Cys-mcMMAF Following IV Dose of GSK2857916 in Participants With Relapsed/Refractory MM- Part 1
Description: Blood samples were collected at designated timepoints. PK parameters of Cys-mcMMAF were calculated using non-compartmental methods. NA indicates that the geometric mean and geometric coefficient of variation could not be calculated since the concentration was not quantifiable.
Time Frame: as for outcome 46
Population: as for outcome 46
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Picograms per milliliter
Arm/Group | Part 1: GSK2857916 0.03 mg/kg | Part 1: GSK2857916 0.06 mg/kg | Part 1: GSK2857916 0.12 mg/kg | Part 1: GSK2857916 0.24 mg/kg | Part 1: GSK2857916 0.48 mg/kg | Part 1: GSK2857916 0.96 mg/kg | Part 1: GSK2857916 1.92 mg/kg | Part 1: GSK2857916 3.40 mg/kg | Part 1: GSK2857916 4.60 mg/kg
Number analyzed (Participants) | 1 | 1 | 4 | 4 | 4 | 3 | 4 | 3 | 6
Picograms per milliliter
  Day 1, Cycle 1,n=0,1,4,2,1,3,3,2,6: number analyzed (Participants) | 0 | 1 | 4 | 2 | 1 | 3 | 3 | 2 | 6
  Day 1, Cycle 1,n=0,1,4,2,1,3,3,2,6 |  | NA (NA) — NA indicates that the geometric mean and geometric coefficient of variation could not be calculated since the concentration was not quantifiable. | NA (NA) — NA indicates that the geometric mean and geometric coefficient of variation could not be calculated since the concentration was not quantifiable. | NA (NA) — NA indicates that the geometric mean and geometric coefficient of variation could not be calculated since the concentration was not quantifiable. | NA (NA) — NA indicates that the geometric mean and geometric coefficient of variation could not be calculated since the concentration was not quantifiable. | NA (NA) — NA indicates that the geometric mean and geometric coefficient of variation could not be calculated since the concentration was not quantifiable. | NA (NA) — NA indicates that the geometric mean and geometric coefficient of variation could not be calculated since the concentration was not quantifiable. | NA (NA) — NA indicates that the geometric mean and geometric coefficient of variation could not be calculated since the concentration was not quantifiable. | NA (NA) — NA indicates that the geometric mean and geometric coefficient of variation could not be calculated since the concentration was not quantifiable.
  Day 1, Cycle 2,n=0,1,0,2,1,2,2,2,5: number analyzed (Participants) | 0 | 1 | 0 | 2 | 1 | 2 | 2 | 2 | 5
  Day 1, Cycle 2,n=0,1,0,2,1,2,2,2,5 |  | NA (NA) — NA indicates that the geometric mean and geometric coefficient of variation could not be calculated since the concentration was not quantifiable. |  | NA (NA) — NA indicates that the geometric mean and geometric coefficient of variation could not be calculated since the concentration was not quantifiable. | NA (NA) — NA indicates that the geometric mean and geometric coefficient of variation could not be calculated since the concentration was not quantifiable. | NA (NA) — NA indicates that the geometric mean and geometric coefficient of variation could not be calculated since the concentration was not quantifiable. | NA (NA) — NA indicates that the geometric mean and geometric coefficient of variation could not be calculated since the concentration was not quantifiable. | NA (NA) — NA indicates that the geometric mean and geometric coefficient of variation could not be calculated since the concentration was not quantifiable. | NA (NA) — NA indicates that the geometric mean and geometric coefficient of variation could not be calculated since the concentration was not quantifiable.
  Day 1, Cycle 4,n=0,0,0,0,0,0,0,0,0: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

61. Secondary Outcome: Ctrough of Cys-mcMMAF Following IV Dose of GSK2857916 in Participants With Relapsed/Refractory MM- Part 1: GSK2857916 2.50 mg/kg
Description: as for outcome 60
Time Frame: Pre-dose and EOI of Day 1 (Cycle 1, Cycle 2 and Cycle 4)
Population: as for outcome 46
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Picograms per milliliter
Arm/Group | Part 1: GSK2857916 2.50 mg/kg
Number analyzed (Participants) | 8
Picograms per milliliter
  Day 1, Cycle 1,n=8 | NA (NA) — NA indicates that the geometric mean and geometric coefficient of variation could not be calculated since the concentration was not quantifiable.
  Day 1, Cycle 2,n=4: number analyzed (Participants) | 4
  Day 1, Cycle 2,n=4 | NA (NA) — NA indicates that the geometric mean and geometric coefficient of variation could not be calculated since the concentration was not quantifiable.
  Day 1, Cycle 4,n=3: number analyzed (Participants) | 3
  Day 1, Cycle 4,n=3 | NA (NA) — NA indicates that the geometric mean and geometric coefficient of variation could not be calculated since the concentration was not quantifiable.

62. Secondary Outcome: Tmax of Cys-mcMMAF Following IV Dose of GSK2857916 in Participants With Relapsed/Refractory MM- Part 1
Description: Blood samples were collected at designated timepoints. PK parameters of Cys-mcMMAF were calculated using non-compartmental methods. Median and full range of Tmax have been presented.
Time Frame: Pre-dose, 30 minutes post-SOI, at EOI, 1, 3, 8 and 24 hours post-EOI of Day 1 (Cycle 1)
Population: PK Part 1 Population. Only those participants with data available at the specified data points were analyzed.
Measure: Median (Full Range); unit: Hours
Arm/Group | Part 1: GSK2857916 0.03 mg/kg | Part 1: GSK2857916 0.06 mg/kg | Part 1: GSK2857916 0.12 mg/kg | Part 1: GSK2857916 0.24 mg/kg | Part 1: GSK2857916 0.48 mg/kg | Part 1: GSK2857916 0.96 mg/kg | Part 1: GSK2857916 1.92 mg/kg | Part 1: GSK2857916 3.40 mg/kg | Part 1: GSK2857916 4.60 mg/kg
Number analyzed (Participants) | 0 | 0 | 1 | 4 | 3 | 3 | 3 | 3 | 6
Hours |  |  | 49.130 [49.13 to 49.13] | 23.875 [9.00 to 24.63] | 24.730 [24.00 to 25.83] | 9.050 [8.78 to 22.83] | 8.750 [7.75 to 24.00] | 23.700 [23.17 to 24.97] | 24.040 [7.83 to 25.00]

63. Secondary Outcome: Tmax of Cys-mcMMAF Following IV Dose of GSK2857916 in Participants With Relapsed/Refractory MM-Part 1: GSK2857916 2.50 mg/kg
Description: as for outcome 62
Time Frame: Pre-dose and EOI of Day 1 (Cycle 1)
Population: PK Part 1 Population. Only those participants with data available at the specified data points were analyzed.
Arm/Group | Part 1: GSK2857916 2.50 mg/kg
Number analyzed (Participants) | 0

64. Secondary Outcome: Number of Participants With at Least One Confirmed Positive Post-Baseline Anti-drug Antibody Result- Part 1
Description: Serum samples were collected for the determination of anti-GSK2857916 antibodies (ADA) using a validated electrochemiluminescent (ECL) immunoassay. The assay involved screening, confirmation and titration steps. If serum samples contained ADA, they were further analyzed for the specificity of antibodies by a confirmation assay. Confirmed positive samples were titrated to obtain the titers of antibodies. The number of participants with at least one confirmed positive ADA at any time post-Baseline is presented.
Time Frame: Up to 21.6 months (maximum duration of follow-up from first dose to last contact or death)
Population: Part 1 Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: GSK2857916 0.03 mg/kg | Part 1: GSK2857916 0.06 mg/kg | Part 1: GSK2857916 0.12 mg/kg | Part 1: GSK2857916 0.24 mg/kg | Part 1: GSK2857916 0.48 mg/kg | Part 1: GSK2857916 0.96 mg/kg | Part 1: GSK2857916 1.92 mg/kg | Part 1: GSK2857916 2.50 mg/kg | Part 1: GSK2857916 3.40 mg/kg | Part 1: GSK2857916 4.60 mg/kg
Number analyzed (Participants) | 1 | 1 | 4 | 4 | 4 | 3 | 4 | 8 | 3 | 6
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

65. Secondary Outcome: Number of Participants With at Least One Confirmed Positive Post-Baseline Anti-drug Antibody Result- Part 2 (MM)
Description: Serum samples were collected for the determination of anti-GSK2857916 antibodies (ADA) using a validated ECL immunoassay. The assay involved screening, confirmation and titration steps. If serum samples contained ADA, they were further analyzed for the specificity of antibodies by a confirmation assay. Confirmed positive samples were titrated to obtain the titers of antibodies. The number of participants with at least one confirmed positive ADA at any time post-Baseline is presented.
Time Frame: Up to 24.2 months (maximum duration of follow-up from first dose to last contact or death)
Population: Part 2 MM Population. Only those participants with data available at the specified data points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: GSK2857916 3.40 mg/kg (MM)
Number analyzed (Participants) | 33
Participants | 0

66. Secondary Outcome: Number of Participants With at Least One Confirmed Positive Post-Baseline Anti-drug Antibody Result- Part 2 (NHL)
Description: Serum samples were collected for the determination of anti-GSK2857916 antibodies (ADA) using a validated ECLimmunoassay. The assay involved screening, confirmation and titration steps. If serum samples contained ADA, they were further analyzed for the specificity of antibodies by a confirmation assay. Confirmed positive samples were titrated to obtain the titers of antibodies. The number of participants with at least one confirmed positive ADA at any time post-Baseline is presented.
Time Frame: Up to 7.2 months (maximum duration of follow-up from first dose to last contact or death)
Population: Part 2 NHL Population. Only those participants with data available at the specified data points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: GSK2857916 3.40 mg/kg (NHL)
Number analyzed (Participants) | 5
Participants | 0

67. Secondary Outcome: Number of Participants With Antibodies to GSK2857916 in Serum Over Time- Part 1
Description: Serum samples were collected for the determination of ADA using a validated ECL immunoassay. The assay involved screening, confirmation and titration steps. If serum samples contained ADA, they were further analyzed for the specificity of antibodies by a confirmation assay. Confirmed positive (pos) samples were titrated to obtain the titers of antibodies. The number of participants with screening, confirming and negative (neg) conclusive ADA results at Baseline and different timepoints is presented.
Time Frame: Baseline, Day 1 (Cycle 2, 3, 4, 6, 9, 12, 16), End of study (within 30 days [+ 7 days of last treatment or prior to the start of new anti-cancer treatment], whichever is earlier) (1 cycle=21 days)
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: GSK2857916 0.03 mg/kg | Part 1: GSK2857916 0.06 mg/kg | Part 1: GSK2857916 0.12 mg/kg | Part 1: GSK2857916 0.24 mg/kg | Part 1: GSK2857916 0.48 mg/kg | Part 1: GSK2857916 0.96 mg/kg | Part 1: GSK2857916 1.92 mg/kg | Part 1: GSK2857916 2.50 mg/kg | Part 1: GSK2857916 3.40 mg/kg | Part 1: GSK2857916 4.60 mg/kg
Number analyzed (Participants) | 1 | 1 | 4 | 4 | 4 | 3 | 4 | 8 | 3 | 6
Participants
  Baseline,screening,pos, n=1,1,4,4,4,3,4,7,2,6: number analyzed (Participants) | 1 | 1 | 4 | 4 | 4 | 3 | 4 | 7 | 2 | 6
  Baseline,screening,pos, n=1,1,4,4,4,3,4,7,2,6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Baseline,screening,neg, n=1,1,4,4,4,3,4,7,2,6: number analyzed (Participants) | 1 | 1 | 4 | 4 | 4 | 3 | 4 | 7 | 2 | 6
  Baseline,screening,neg, n=1,1,4,4,4,3,4,7,2,6 | 1 | 1 | 4 | 4 | 4 | 3 | 4 | 7 | 2 | 6
  Baseline,confirming,pos,n=0,0,0,0,0,0,0,0,0,0: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Baseline,confirming,neg,n=0,0,0,0,0,0,0,0,0,0: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Baseline,neg,conclusive,n=1,1,4,4,4,3,4,7,2,6: number analyzed (Participants) | 1 | 1 | 4 | 4 | 4 | 3 | 4 | 7 | 2 | 6
  Baseline,neg,conclusive,n=1,1,4,4,4,3,4,7,2,6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 0 | 0
  Cycle 2 Day 1,screening,pos, n=0,1,4,2,2,3,3,8,3,5: number analyzed (Participants) | 0 | 1 | 4 | 2 | 2 | 3 | 3 | 8 | 3 | 5
  Cycle 2 Day 1,screening,pos, n=0,1,4,2,2,3,3,8,3,5 |  | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Cycle 2 Day 1,screening,neg, n=0,1,4,2,2,3,3,8,3,5: number analyzed (Participants) | 0 | 1 | 4 | 2 | 2 | 3 | 3 | 8 | 3 | 5
  Cycle 2 Day 1,screening,neg, n=0,1,4,2,2,3,3,8,3,5 |  | 1 | 4 | 2 | 2 | 3 | 3 | 8 | 3 | 5
  Cycle 2 Day 1,confirming,pos,n=0,0,0,0,0,0,0,0,0,0: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Cycle 2 Day 1,confirming,neg,n=0,0,0,0,0,0,0,0,0,0: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Cycle 2 Day 1,neg,conclusive,n=0,1,4,2,2,3,3,8,3,5: number analyzed (Participants) | 0 | 1 | 4 | 2 | 2 | 3 | 3 | 8 | 3 | 5
  Cycle 2 Day 1,neg,conclusive,n=0,1,4,2,2,3,3,8,3,5 |  | 1 | 3 | 2 | 2 | 3 | 3 | 8 | 2 | 5
  Cycle 3 Day 1,screening,pos, n=0,1,0,2,2,1,2,4,3,6: number analyzed (Participants) | 0 | 1 | 0 | 2 | 2 | 1 | 2 | 4 | 3 | 6
  Cycle 3 Day 1,screening,pos, n=0,1,0,2,2,1,2,4,3,6 |  | 0 |  | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Cycle 3 Day 1,screening,neg, n=0,1,0,2,2,1,2,4,3,6: number analyzed (Participants) | 0 | 1 | 0 | 2 | 2 | 1 | 2 | 4 | 3 | 6
  Cycle 3 Day 1,screening,neg, n=0,1,0,2,2,1,2,4,3,6 |  | 1 |  | 2 | 2 | 1 | 2 | 4 | 3 | 6
  Cycle 3 Day 1,confirming,pos,n=0,0,0,0,0,0,0,0,0,0: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Cycle 3 Day 1,confirming,neg,n=0,0,0,0,0,0,0,0,0,0: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Cycle 3 Day 1,neg,conclusive,n=0,1,0,2,2,1,2,4,3,6: number analyzed (Participants) | 0 | 1 | 0 | 2 | 2 | 1 | 2 | 4 | 3 | 6
  Cycle 3 Day 1,neg,conclusive,n=0,1,0,2,2,1,2,4,3,6 |  | 1 |  | 2 | 2 | 1 | 2 | 2 | 0 | 4
  Cycle 4 Day 1,screening,pos, n=0,0,0,0,0,0,0,0,0,1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Cycle 4 Day 1,screening,pos, n=0,0,0,0,0,0,0,0,0,1 |  |  |  |  |  |  |  |  |  | 0
  Cycle 4 Day 1,screening,neg, n=0,0,0,0,0,0,0,0,0,1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Cycle 4 Day 1,screening,neg, n=0,0,0,0,0,0,0,0,0,1 |  |  |  |  |  |  |  |  |  | 1
  Cycle 4 Day 1,confirming,pos,n=0,0,0,0,0,0,0,0,0,0: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Cycle 4 Day 1,confirming,neg,n=0,0,0,0,0,0,0,0,0,0: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Cycle 4 Day 1,neg,conclusive,n=0,0,0,0,0,0,0,0,0,1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Cycle 4 Day 1,neg,conclusive,n=0,0,0,0,0,0,0,0,0,1 |  |  |  |  |  |  |  |  |  | 0
  Cycle 6 Day 1,screening,pos, n=0,0,0,1,1,1,2,3,3,3: number analyzed (Participants) | 0 | 0 | 0 | 1 | 1 | 1 | 2 | 3 | 3 | 3
  Cycle 6 Day 1,screening,pos, n=0,0,0,1,1,1,2,3,3,3 |  |  |  | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Cycle 6 Day 1,screening,neg, n=0,0,0,1,1,1,2,3,3,3: number analyzed (Participants) | 0 | 0 | 0 | 1 | 1 | 1 | 2 | 3 | 3 | 3
  Cycle 6 Day 1,screening,neg, n=0,0,0,1,1,1,2,3,3,3 |  |  |  | 1 | 1 | 1 | 2 | 3 | 2 | 3
  Cycle 6 Day 1,confirming,pos,n=0,0,0,0,0,0,0,0,1,0: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Cycle 6 Day 1,confirming,pos,n=0,0,0,0,0,0,0,0,1,0 |  |  |  |  |  |  |  |  | 0 |
  Cycle 6 Day 1,confirming,neg,n=0,0,0,0,0,0,0,0,1,0: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Cycle 6 Day 1,confirming,neg,n=0,0,0,0,0,0,0,0,1,0 |  |  |  |  |  |  |  |  | 1 |
  Cycle 6 Day 1,neg,conclusive,n=0,0,0,1,1,1,2,3,3,3: number analyzed (Participants) | 0 | 0 | 0 | 1 | 1 | 1 | 2 | 3 | 3 | 3
  Cycle 6 Day 1,neg,conclusive,n=0,0,0,1,1,1,2,3,3,3 |  |  |  | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Cycle 9 Day 1,screening,pos, n=0,0,0,1,0,0,1,1,2,2: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 2 | 2
  Cycle 9 Day 1,screening,pos, n=0,0,0,1,0,0,1,1,2,2 |  |  |  | 0 |  |  | 0 | 0 | 0 | 0
  Cycle 9 Day 1,screening,neg, n=0,0,0,1,0,0,1,1,2,2: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 2 | 2
  Cycle 9 Day 1,screening,neg, n=0,0,0,1,0,0,1,1,2,2 |  |  |  | 1 |  |  | 1 | 1 | 2 | 2
  Cycle 9 Day 1,confirming,pos,n=0,0,0,0,0,0,0,0,0,0: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Cycle 9 Day 1,confirming,neg,n=0,0,0,0,0,0,0,0,0,0: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Cycle 9 Day 1,neg,conclusive,n=0,0,0,1,0,0,1,1,2,2: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 2 | 2
  Cycle 9 Day 1,neg,conclusive,n=0,0,0,1,0,0,1,1,2,2 |  |  |  | 0 |  |  | 0 | 0 | 0 | 0
  Cycle 12 Day 1,screening,pos,n=0,0,0,1,0,0,1,1,1,3: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 3
  Cycle 12 Day 1,screening,pos,n=0,0,0,1,0,0,1,1,1,3 |  |  |  | 0 |  |  | 0 | 0 | 0 | 1
  Cycle 12 Day 1,screening,neg,n=0,0,0,1,0,0,1,1,1,3: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 3
  Cycle 12 Day 1,screening,neg,n=0,0,0,1,0,0,1,1,1,3 |  |  |  | 1 |  |  | 1 | 1 | 1 | 2
  Cycle 12 Day1,confirming,pos,n=0,0,0,0,0,0,0,0,0,1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Cycle 12 Day1,confirming,pos,n=0,0,0,0,0,0,0,0,0,1 |  |  |  |  |  |  |  |  |  | 0
  Cycle 12 Day1,confirming,neg,n=0,0,0,0,0,0,0,0,0,1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Cycle 12 Day1,confirming,neg,n=0,0,0,0,0,0,0,0,0,1 |  |  |  |  |  |  |  |  |  | 1
  Cycle 12 Day1,neg,conclusive,n=0,0,0,1,0,0,1,1,1,3: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 3
  Cycle 12 Day1,neg,conclusive,n=0,0,0,1,0,0,1,1,1,3 |  |  |  | 0 |  |  | 0 | 0 | 0 | 0
  Cycle 16 Day 1,screening,pos,n=0,0,0,0,0,0,1,1,1,2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 2
  Cycle 16 Day 1,screening,pos,n=0,0,0,0,0,0,1,1,1,2 |  |  |  |  |  |  | 0 | 0 | 0 | 0
  Cycle 16 Day 1,screening,neg,n=0,0,0,0,0,0,1,1,1,2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 2
  Cycle 16 Day 1,screening,neg,n=0,0,0,0,0,0,1,1,1,2 |  |  |  |  |  |  | 1 | 1 | 1 | 2
  Cycle 16 Day1,confirming,pos,n=0,0,0,0,0,0,0,0,0,0: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Cycle 16 Day1,confirming,neg,n=0,0,0,0,0,0,0,0,0,0: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Cycle 16 Day1,neg,conclusive,n=0,0,0,0,0,0,1,1,1,2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 2
  Cycle 16 Day1,neg,conclusive,n=0,0,0,0,0,0,1,1,1,2 |  |  |  |  |  |  | 0 | 0 | 0 | 0
  End of study,screening,pos,n=1,1,4,4,4,3,3,6,1,5: number analyzed (Participants) | 1 | 1 | 4 | 4 | 4 | 3 | 3 | 6 | 1 | 5
  End of study,screening,pos,n=1,1,4,4,4,3,3,6,1,5 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  End of study,screening,neg,n=1,1,4,4,4,3,3,6,1,5: number analyzed (Participants) | 1 | 1 | 4 | 4 | 4 | 3 | 3 | 6 | 1 | 5
  End of study,screening,neg,n=1,1,4,4,4,3,3,6,1,5 | 1 | 1 | 4 | 3 | 4 | 3 | 3 | 6 | 1 | 5
  End of study,confirming,pos,n=0,0,0,1,0,0,0,0,0,0: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  End of study,confirming,pos,n=0,0,0,1,0,0,0,0,0,0 |  |  |  | 0 |  |  |  |  |  |
  End of study,confirming,neg,n=0,0,0,1,0,0,0,0,0,0: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  End of study,confirming,neg,n=0,0,0,1,0,0,0,0,0,0 |  |  |  | 1 |  |  |  |  |  |
  End of study,neg,conclusive,n=1,1,4,4,4,3,3,6,1,5: number analyzed (Participants) | 1 | 1 | 4 | 4 | 4 | 3 | 3 | 6 | 1 | 5
  End of study,neg,conclusive,n=1,1,4,4,4,3,3,6,1,5 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

68. Secondary Outcome: Number of Participants With Antibodies to GSK2857916 in Serum Over Time- Part 2 (MM)
Description: Serum samples were collected for the determination of ADA using a validated ECL immunoassay. The assay involved screening, confirmation and titration steps. If serum samples contained ADA, they were further analyzed for the specificity of antibodies by a confirmation assay. Confirmed positive samples were titrated to obtain the titers of antibodies. The number of participants with screening, confirming and negative conclusive ADA results at Baseline and different timepoints is presented.
Time Frame: Baseline, Day 1 (Cycle 2, 3, 6, 7, 9, 11, 12, 16), End of study (within 30 days [+ 7 days of last treatment or prior to the start of new anti-cancer treatment], whichever is earlier) (1 cycle=21 days)
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: GSK2857916 3.40 mg/kg (MM)
Number analyzed (Participants) | 35
Participants
  Baseline, screening, positive, n=30: number analyzed (Participants) | 30
  Baseline, screening, positive, n=30 | 2
  Baseline, screening, negative n=30: number analyzed (Participants) | 30
  Baseline, screening, negative n=30 | 28
  Baseline, confirming, positive, n=2: number analyzed (Participants) | 2
  Baseline, confirming, positive, n=2 | 0
  Baseline, confirming, negative, n=2: number analyzed (Participants) | 2
  Baseline, confirming, negative, n=2 | 2
  Baseline, negative, conclusive, n=30: number analyzed (Participants) | 30
  Baseline, negative, conclusive, n=30 | 21
  Cycle 2, Day 1, screening, positive, n=31: number analyzed (Participants) | 31
  Cycle 2, Day 1, screening, positive, n=31 | 3
  Cycle 2, Day 1, screening, negative, n=31: number analyzed (Participants) | 31
  Cycle 2, Day 1, screening, negative, n=31 | 28
  Cycle 2, Day 1, confirming, positive, n=3: number analyzed (Participants) | 3
  Cycle 2, Day 1, confirming, positive, n=3 | 0
  Cycle 2, Day 1, confirming, negative, n=3: number analyzed (Participants) | 3
  Cycle 2, Day 1, confirming, negative, n=3 | 3
  Cycle 2, Day 1, negative, conclusive, n=31: number analyzed (Participants) | 31
  Cycle 2, Day 1, negative, conclusive, n=31 | 27
  Cycle 3, Day 1, screening, positive, n=23: number analyzed (Participants) | 23
  Cycle 3, Day 1, screening, positive, n=23 | 0
  Cycle 3, Day 1, screening, negative, n=23: number analyzed (Participants) | 23
  Cycle 3, Day 1, screening, negative, n=23 | 23
  Cycle 3, Day 1, confirming, positive, n=0: number analyzed (Participants) | 0
  Cycle 3, Day 1, confirming, negative, n=0: number analyzed (Participants) | 0
  Cycle 3, Day 1, negative, conclusive, n=23: number analyzed (Participants) | 23
  Cycle 3, Day 1, negative, conclusive, n=23 | 14
  Cycle 6, Day 1, screening, positive, n=17: number analyzed (Participants) | 17
  Cycle 6, Day 1, screening, positive, n=17 | 4
  Cycle 6, Day 1, screening, negative, n=17: number analyzed (Participants) | 17
  Cycle 6, Day 1, screening, negative, n=17 | 13
  Cycle 6, Day 1, confirming, positive, n=4: number analyzed (Participants) | 4
  Cycle 6, Day 1, confirming, positive, n=4 | 0
  Cycle 6, Day 1, confirming, negative, n=4: number analyzed (Participants) | 4
  Cycle 6, Day 1, confirming, negative, n=4 | 4
  Cycle 6, Day 1, negative, conclusive, n=17: number analyzed (Participants) | 17
  Cycle 6, Day 1, negative, conclusive, n=17 | 0
  Cycle 7, Day 1, screening, positive, n=1: number analyzed (Participants) | 1
  Cycle 7, Day 1, screening, positive, n=1 | 0
  Cycle 7, Day 1, screening, negative, n=1: number analyzed (Participants) | 1
  Cycle 7, Day 1, screening, negative, n=1 | 1
  Cycle 7, Day 1, confirming, positive, n=0: number analyzed (Participants) | 0
  Cycle 7, Day 1, confirming, negative, n=0: number analyzed (Participants) | 0
  Cycle 7, Day 1, negative, conclusive, n=1: number analyzed (Participants) | 1
  Cycle 7, Day 1, negative, conclusive, n=1 | 0
  Cycle 9, Day 1, screening, positive, n=16: number analyzed (Participants) | 16
  Cycle 9, Day 1, screening, positive, n=16 | 2
  Cycle 9, Day 1, screening, negative, n=16: number analyzed (Participants) | 16
  Cycle 9, Day 1, screening, negative, n=16 | 14
  Cycle 9, Day 1, confirming, positive, n=2: number analyzed (Participants) | 2
  Cycle 9, Day 1, confirming, positive, n=2 | 0
  Cycle 9, Day 1, confirming, negative, n=2: number analyzed (Participants) | 2
  Cycle 9, Day 1, confirming, negative, n=2 | 2
  Cycle 9, Day 1, negative, conclusive, n=16: number analyzed (Participants) | 16
  Cycle 9, Day 1, negative, conclusive, n=16 | 0
  Cycle 11, Day 1, screening, positive, n=1: number analyzed (Participants) | 1
  Cycle 11, Day 1, screening, positive, n=1 | 0
  Cycle 11, Day 1, screening, negative, n=1: number analyzed (Participants) | 1
  Cycle 11, Day 1, screening, negative, n=1 | 1
  Cycle 11, Day 1, confirming, positive, n=0: number analyzed (Participants) | 0
  Cycle 11, Day 1, confirming, negative, n=0: number analyzed (Participants) | 0
  Cycle 11, Day 1, negative, conclusive, n=1: number analyzed (Participants) | 1
  Cycle 11, Day 1, negative, conclusive, n=1 | 0
  Cycle 12, Day 1, screening, positive, n=8: number analyzed (Participants) | 8
  Cycle 12, Day 1, screening, positive, n=8 | 0
  Cycle 12, Day 1, screening, negative, n=8: number analyzed (Participants) | 8
  Cycle 12, Day 1, screening, negative, n=8 | 8
  Cycle 12, Day 1, confirming, positive, n=0: number analyzed (Participants) | 0
  Cycle 12, Day 1, confirming, negative, n=0: number analyzed (Participants) | 0
  Cycle 12, Day 1, negative, conclusive, n=8: number analyzed (Participants) | 8
  Cycle 12, Day 1, negative, conclusive, n=8 | 0
  Cycle 16, Day 1, screening, positive, n=8: number analyzed (Participants) | 8
  Cycle 16, Day 1, screening, positive, n=8 | 0
  Cycle 16, Day 1, screening, negative, n=8: number analyzed (Participants) | 8
  Cycle 16, Day 1, screening, negative, n=8 | 8
  Cycle 16, Day 1, confirming, positive, n=0: number analyzed (Participants) | 0
  Cycle 16, Day 1, confirming, negative, n=0: number analyzed (Participants) | 0
  Cycle 16, Day 1, negative, conclusive, n=8: number analyzed (Participants) | 8
  Cycle 16, Day 1, negative, conclusive, n=8 | 0
  End of study, screening, positive, n=21: number analyzed (Participants) | 21
  End of study, screening, positive, n=21 | 1
  End of study, screening, negative, n=21: number analyzed (Participants) | 21
  End of study, screening, negative, n=21 | 20
  End of study, confirming, positive, n=1: number analyzed (Participants) | 1
  End of study, confirming, positive, n=1 | 0
  End of study, confirming, negative, n=1: number analyzed (Participants) | 1
  End of study, confirming, negative, n=1 | 1
  End of study, negative, conclusive, n=21: number analyzed (Participants) | 21
  End of study, negative, conclusive, n=21 | 0

69. Secondary Outcome: Number of Participants With Antibodies to GSK2857916 in Serum Over Time - Part 2 (NHL)
Description: as for outcome 68
Time Frame: Baseline, Day 1 (Cycle 2, 3), End of study (within 30 days [+ 7 days of last treatment or prior to the start of new anti-cancer treatment], whichever is earlier) (1 cycle=21 days)
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: GSK2857916 3.40 mg/kg (NHL)
Number analyzed (Participants) | 5
Participants
  Baseline, screening, positive, n=5 | 0
  Baseline, screening, negative n=5 | 5
  Baseline, confirming, positive, n=0: number analyzed (Participants) | 0
  Baseline, confirming, negative, n=0: number analyzed (Participants) | 0
  Baseline, negative, conclusive, n=5 | 5
  Cycle 2, Day 1, screening, positive, n=4: number analyzed (Participants) | 4
  Cycle 2, Day 1, screening, positive, n=4 | 0
  Cycle 2, Day 1, screening, negative, n=4: number analyzed (Participants) | 4
  Cycle 2, Day 1, screening, negative, n=4 | 4
  Cycle 2, Day 1, confirming, positive, n=0: number analyzed (Participants) | 0
  Cycle 2, Day 1, confirming, negative, n=0: number analyzed (Participants) | 0
  Cycle 2, Day 1, negative, conclusive, n=4: number analyzed (Participants) | 4
  Cycle 2, Day 1, negative, conclusive, n=4 | 4
  Cycle 3, Day 1, screening, positive, n=2: number analyzed (Participants) | 2
  Cycle 3, Day 1, screening, positive, n=2 | 1
  Cycle 3, Day 1, screening, negative, n=2: number analyzed (Participants) | 2
  Cycle 3, Day 1, screening, negative, n=2 | 1
  Cycle 3, Day 1, confirming, positive, n=1: number analyzed (Participants) | 1
  Cycle 3, Day 1, confirming, positive, n=1 | 0
  Cycle 3, Day 1, confirming, negative, n=1: number analyzed (Participants) | 1
  Cycle 3, Day 1, confirming, negative, n=1 | 1
  Cycle 3, Day 1, negative, conclusive, n=2: number analyzed (Participants) | 2
  Cycle 3, Day 1, negative, conclusive, n=2 | 1
  End of study, screening, positive, n=4: number analyzed (Participants) | 4
  End of study, screening, positive, n=4 | 0
  End of study, screening, negative, n=4: number analyzed (Participants) | 4
  End of study, screening, negative, n=4 | 4
  End of study, confirming, positive, n=0: number analyzed (Participants) | 0
  End of study, confirming, negative, n=0: number analyzed (Participants) | 0
  End of study, negative, conclusive, n=4: number analyzed (Participants) | 4
  End of study, negative, conclusive, n=4 | 0

70. Secondary Outcome: Overall Response Rate (ORR)- Part 1
Description: ORR was determined by the investigator according to international myeloma working group uniform response criteria for MM (IMWG 2011). ORR was calculated as the number of participants with best overall response of stringent complete response (sCR), complete response (CR), very good partial response (VGPR) and partial response (PR).
Time Frame: From the Start of Treatment (at First Dose) up to the earlier of disease progression or the start of new anti-cancer therapy (maximum duration of follow-up is 21.6 months)
Population: Part 1 Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: GSK2857916 0.03 mg/kg | Part 1: GSK2857916 0.06 mg/kg | Part 1: GSK2857916 0.12 mg/kg | Part 1: GSK2857916 0.24 mg/kg | Part 1: GSK2857916 0.48 mg/kg | Part 1: GSK2857916 0.96 mg/kg | Part 1: GSK2857916 1.92 mg/kg | Part 1: GSK2857916 2.50 mg/kg | Part 1: GSK2857916 3.40 mg/kg | Part 1: GSK2857916 4.60 mg/kg
Number analyzed (Participants) | 1 | 1 | 4 | 4 | 4 | 3 | 4 | 8 | 3 | 6
Participants | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 3 | 3

71. Secondary Outcome: ORR-Part 2 (MM)
Description: ORR was determined by the investigator according to IMWG 2011 uniform response criteria for MM. ORR was calculated as the number of participants with best overall response of sCR, CR, VGPR and PR.
Time Frame: From the Start of Treatment (at First Dose) up to the earlier of disease progression or the start of new anti-cancer therapy (maximum duration of follow-up is 24.2 months)
Population: Part 2 MM Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: GSK2857916 3.40 mg/kg (MM)
Number analyzed (Participants) | 35
Participants | 21

72. Secondary Outcome: ORR-Part 2 (NHL)
Description: Overall Response Rate in NHL population was determined by the investigator according to Revised Response Criteria for Malignant Lymphoma. ORR was calculated as the number of participants with confirmed complete remission (CR) or partial remission (PR). Complete remission was defined as disappearance of all evidence of disease and partial remission was defined as regression of measurable disease and no new sites.
Time Frame: From the Start of Treatment (at First Dose) up to the earlier of disease progression or the start of new anti-cancer therapy (maximum duration of follow-up is 7.2 months)
Population: Part 2 NHL Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: GSK2857916 3.40 mg/kg (NHL)
Number analyzed (Participants) | 6
Participants | 0

73. Secondary Outcome: Clinical Benefit Rate (CBR)- Part 1
Description: CBR was calculated as the number of participants with best overall response of sCR, CR, VGPR, PR and minimal response (MR).
Time Frame: as for outcome 70
Population: Part 1 Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: GSK2857916 0.03 mg/kg | Part 1: GSK2857916 0.06 mg/kg | Part 1: GSK2857916 0.12 mg/kg | Part 1: GSK2857916 0.24 mg/kg | Part 1: GSK2857916 0.48 mg/kg | Part 1: GSK2857916 0.96 mg/kg | Part 1: GSK2857916 1.92 mg/kg | Part 1: GSK2857916 2.50 mg/kg | Part 1: GSK2857916 3.40 mg/kg | Part 1: GSK2857916 4.60 mg/kg
Number analyzed (Participants) | 1 | 1 | 4 | 4 | 4 | 3 | 4 | 8 | 3 | 6
Participants | 0 | 0 | 0 | 1 | 1 | 1 | 2 | 2 | 3 | 5

74. Secondary Outcome: CBR- Part 2
Description: CBR was calculated as the number of participants with best overall response of sCR, CR, VGPR, PR and MR.
Time Frame: as for outcome 71
Population: Part 2 MM Population. Data is presented only for Part 2 MM Population; since this analysis was not planned for Part 2 NHL Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: GSK2857916 3.40 mg/kg (MM)
Number analyzed (Participants) | 35
Participants | 21

ADVERSE EVENTS:
Time Frame: SAEs & common (>=5%) non-SAEs were collected from start of study treatment until 23.5 months for Part 1, 35 months for Part 2 (MM) and 7.2 months for Part 2 (NHL)
Description: SAEs and common (>=5%) non-SAEs were reported by treatment for the Part 1 Population which comprised of all Part 1 participants (exclusively MM) who received at least one dose of GSK2857916; Part 2 MM and NHL Population which comprised of all Part 2 MM and NHL participants who received at least one dose of GSK2857916.
Arm/Group | Part 1: GSK2857916 0.03 mg/kg | Part 1: GSK2857916 0.06 mg/kg | Part 1: GSK2857916 0.12 mg/kg | Part 1: GSK2857916 0.24 mg/kg | Part 1: GSK2857916 0.48 mg/kg | Part 1: GSK2857916 0.96 mg/kg | Part 1: GSK2857916 1.92 mg/kg | Part 1: GSK2857916 2.50 mg/kg | Part 1: GSK2857916 3.40 mg/kg | Part 1: GSK2857916 4.60 mg/kg | Part 2: GSK2857916 3.40 mg/kg (MM) | Part 2: GSK2857916 3.40 mg/kg (NHL)
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/1 | 0/4 | 0/4 | 0/4 | 0/3 | 0/4 | 1/8 | 0/3 | 1/6 | 5/35 | 3/6
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/1 | 1/4 | 1/4 | 1/4 | 0/3 | 2/4 | 4/8 | 1/3 | 3/6 | 17/35 | 3/6
Other Adverse Events (participants affected / at risk) | 1/1 | 1/1 | 4/4 | 4/4 | 3/4 | 3/3 | 4/4 | 8/8 | 3/3 | 6/6 | 35/35 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: GSK2857916 0.03 mg/kg (N=1) | Part 1: GSK2857916 0.06 mg/kg (N=1) | Part 1: GSK2857916 0.12 mg/kg (N=4) | Part 1: GSK2857916 0.24 mg/kg (N=4) | Part 1: GSK2857916 0.48 mg/kg (N=4) | Part 1: GSK2857916 0.96 mg/kg (N=3) | Part 1: GSK2857916 1.92 mg/kg (N=4) | Part 1: GSK2857916 2.50 mg/kg (N=8) | Part 1: GSK2857916 3.40 mg/kg (N=3) | Part 1: GSK2857916 4.60 mg/kg (N=6) | Part 2: GSK2857916 3.40 mg/kg (MM) (N=35) | Part 2: GSK2857916 3.40 mg/kg (NHL) (N=6)
Adenovirus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Babesiosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis infective (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis salmonella (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hyperviscosity syndrome (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Limbal stem cell deficiency (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pharyngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 5 (5) | 0 (0)
Pneumonia haemophilus (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Retinal detachment (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Salmonellosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Spinal cord compression (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: GSK2857916 0.03 mg/kg (N=1) | Part 1: GSK2857916 0.06 mg/kg (N=1) | Part 1: GSK2857916 0.12 mg/kg (N=4) | Part 1: GSK2857916 0.24 mg/kg (N=4) | Part 1: GSK2857916 0.48 mg/kg (N=4) | Part 1: GSK2857916 0.96 mg/kg (N=3) | Part 1: GSK2857916 1.92 mg/kg (N=4) | Part 1: GSK2857916 2.50 mg/kg (N=8) | Part 1: GSK2857916 3.40 mg/kg (N=3) | Part 1: GSK2857916 4.60 mg/kg (N=6) | Part 2: GSK2857916 3.40 mg/kg (MM) (N=35) | Part 2: GSK2857916 3.40 mg/kg (NHL) (N=6)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 7 (8) | 0 (0)
Albuminuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alpha haemolytic streptococcal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 2 (4) | 1 (1) | 3 (3) | 0 (0) | 3 (4) | 10 (12) | 1 (1)
Angina bullosa haemorrhagica (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (4) | 1 (1) | 0 (0) | 1 (1) | 4 (5) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (3) | 4 (5) | 13 (17) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atrial flutter (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Babesiosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 7 (7) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 5 (7) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 3 (3) | 1 (1)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (4) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Borderline glaucoma (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bundle branch block left (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bundle branch block right (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Catheter site discharge (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 2 (2) | 1 (1) | 9 (10) | 1 (1)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Conjunctivitis viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 7 (8) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 5 (5) | 0 (0)
Corneal deposits (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Corneal disorder (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Corneal irritation (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Corneal oedema (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Corneal opacity (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 2 (3) | 0 (0) | 14 (16) | 1 (1)
Cushingoid (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 5 (6) | 0 (0)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 10 (11) | 1 (1)
Diplopia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Disturbance in attention (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 1 (1) | 2 (3) | 1 (1) | 13 (18) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Taste disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6 (6) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Embolism (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 3 (4) | 0 (0)
Eye pain (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 4 (4) | 1 (1)
Eye pruritus (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Facial nerve disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Facial pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 1 (3) | 2 (3) | 1 (1) | 3 (4) | 2 (2) | 4 (4) | 8 (9) | 1 (1)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Foreign body sensation in eyes (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 7 (11) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Gingival bleeding (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (3) | 2 (2) | 5 (5) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Hypercreatininaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 4 (10) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoaesthesia oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 4 (5) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Hypophagia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Increased tendency to bruise (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Intraocular pressure increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 4 (4) | 0 (0)
Keratitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Keratopathy (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lacrimation increased (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (6) | 0 (0)
Lip pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower respiratory tract infection bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (8) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Micturition urgency (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 1 (1) | 4 (4) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 3 (4) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 3 (3) | 3 (3) | 2 (5) | 4 (4) | 11 (15) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 1 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (3) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (5) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nocturia (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ocular hypertension (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ocular toxicity (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0)
Optic disc haemorrhage (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (4) | 0 (0)
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 4 (4) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Photophobia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (3) | 2 (2) | 10 (11) | 0 (0)
Photopsia (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 13 (30) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 4 (5) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Punctate keratitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 2 (3) | 9 (13) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 4 (5) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Restless legs syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 5 (8) | 0 (0)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Spinal cord injury thoracic (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Telangiectasia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (7) | 0 (0) | 1 (1) | 1 (1) | 2 (4) | 5 (9) | 9 (18) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 9 (12) | 0 (0)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 4 (7) | 0 (0)
Urinary tract pain (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 2 (2) | 3 (11) | 4 (4) | 18 (53) | 2 (3)
Visual impairment (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 2 (3) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood immunoglobulin G decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Periorbital swelling (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Jaundice (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2017-11-02): https://cdn.clinicaltrials.gov/large-docs/87/NCT02064387/Prot_000.pdf
  • Statistical Analysis Plan (2019-11-18): https://cdn.clinicaltrials.gov/large-docs/87/NCT02064387/SAP_002.pdf